



August 19, 2020

Martha Kruhm, MS RAC Head, Protocol and Information Office Quality Assurance Section CTEP, DCT, NCI 6130 Executive Blvd, EPN Room 7000 Bethesda, MD 20892

Dear Ms. Kruhm:

Enclosed is Addendum #25 to EAY131-S2, Phase II Study of Trametinib in Patients with Tumors with GNAQ or GNA11 Mutations

This addendum is in response to Dr. Helen Chen's Request for Rapid Amendment for Trametinib dimethyl sulfoxide dated November 19, 2019, and also, Dr. Tali Johnson's Amendment Request for updates to specific protocol language for Trametinib dimethyl sulfoxide dated June 5, 2020

Please replace your current copy of the protocol and Informed Consent document with these updated versions. We recommend that each institution maintain a file containing the original protocol, Informed Consent, and all subsequent revisions/versions.

# **IRB Review Requirements:**

This addendum has been reviewed and approved by the Central IRB, which is the sole IRB of record for this study. Local IRB review and approval is unnecessary.

**Implementation of this addendum must occur on the activation date.** Sites are not permitted to conduct the study utilizing outdated versions of any MATCH protocol documents after the activation date of this addendum.

**Re:** Review of Amendment #36 of Protocol #EAY131-S2: "MATCH Treatment Subprotocol S2: Phase II Study of Trametinib in Patients with Tumors with GNAQ or GNA11 Mutations." The following are ECOG-ACRIN's responses to the CTEP review comments dated 5/26/2020. Please note that the Principal Investigator's comments appear in bold below.

# I. Comments Requiring a Response – Administrative & Editorial Issues:

| # | Section | Comments |
|---|---|---|
| | | This protocol amendment has not completely updated the subprotocol chair's contact information according to CTEP's records. |
| | | Our records indicate: |
| 1. | Title page | <ul> <li>Jason Luke, MD (IVR – 47003) has relocated to University of Pittsburgh<br/>Cancer Institute. Please update his practice site including address.</li> </ul> |
| | | PI Response: Dr. Luke's contact information, including the practice site address, has been updated. |

# II. Additional Protocol Changes by Principal Investigator:

The following revisions to EAY131-S2 protocol have been made in this addendum:

| | Section | Change |
|---|---|---|
| 1. | Cover Page | Updated version date and addendum number. |
| 2. | 3.2.1 | In second box, under "Pregnancies" revised language referencing "subject" to "female patient". |
| 3. | 3.3 | Updated CAEPR list for Trametinib dimethyl sulfoxide with Version 2.6 October 10, 2019 |
| 4. | <u>5</u> | Updated Trametinib dimethyl sulfoxide supply language. |
| 5. | Appendix IV | Updated patient drug information template format. |

The following revisions to EAY131-S2 Informed Consent Document have been made in this addendum:

| | Section | Change |
|---|---|---|
| 1. | Page 1 | Updated version date. |
| 2. | What possible risks can I expect from taking part in this study? | Updated condensed risk list for Trametinib dimethyl sulfoxide with Version 2.6 October 10, 2019. |

If you have any questions regarding this addendum, please contact <a href="mage-agu@ecog-acrin.org">aagu@ecog-acrin.org</a> or 857-504-2900.

We request review and approval of this addendum to EAY131-S2 so ECOG-ACRIN may activate it promptly.

Thank you.

Sincerely,

Pamela Cogliano

Senior Director of Protocol Development



# Molecular Analysis for Therapy Choice (MATCH)

# MATCH Treatment Subprotocol S2: Phase II Study of Trametinib in Patients with Tumors with GNAQ or GNA11 Mutations

TRAMETINIB TREATMENT

SUBPROTOCOL CHAIR: Jason Luke, MD, FACP

TRAMETINIB TREATMENT

SUBPROTOCOL CO-CHAIR: Hussein Tawbi, MD, PhD TRAMETINIB TRANSLATIONAL CHAIR: Andrew Chi, MD, PhD

Version Date: August 19, 2020

NOTE: This subprotocol (EAY131-S2)

should be used in conjunction with

the MATCH Master Protocol

(EAY131)

Rev.5/16

Rev. Add13

Rev. Add19 NOTE: As of 11/17, all protocol changes will

be noted by addendum number.

SUBPROTOCOL ACTIVATION DATE

February 25, 2016 (Incorporated in Addendum

#2)

Addendum #3 – 5/16

Addendum #5 - 12/16

Addendum #6 - 1/17

Addendum #7 - 3/17

Addendum #13

Addendum #19

Addendum #25

| Agent | IND# | NSC# | Supply |
|---|---|---|---|
| Trametinib dimethyl sulfoxide | IND Sponsor: DCTD, NCI IND#: | 763093 | NCI Supplied |

# **Table of Contents**

| Molecular Analysis for Therapy Choice (MATCH) | i |
|---|---|
| MATCH Treatment Subprotocol S2: Phase II Study of Trametinib in Patients | |
| Tumors with GNAQ or GNA11 Mutations | <u>1</u> |
| Table of Contents | 2 |
| Schema | 4 |
| 1. Introduction | 5 |
| 1.1 Trametinib Dimethyl Sulfoxide (GSK1120212B, MEKINIST) | 5 |
| 1.2 Supporting Preliminary Data | 10 |
| 2. Selection of Patients | 13 |
| 2.1 Eligibility Criteria: | 13 |
| 3. Treatment Plan | 15 |
| 3.1 Administration Schedule | 15 |
| 3.2 Adverse Event Reporting Requirements | 15 |
| 3.3 Comprehensive Adverse Events and Potential Risks List (CAEPR) f | or |
| Trametinib dimethyl sulfoxide (GSK1120212B, NSC 763093) | 19 |
| 3.4 Dose Modifications | |
| 3.5 Dose Modifications for Trametinib and supportive care | |
| 3.6 Supportive Care | |
| 3.7 Duration of Agent-specific treatment | |
| 3.8 Duration of Follow-Up | |
| 4. Study Parameters | |
| 4.1 Therapeutic Parameters for Trametinib Treatment | |
| 5. Drug Formulation and Procurement | |
| 5.1 Trametinib dimethyl sulfoxide (NSC 763093) | 40 |
| 6. Translational Studies | 42 |
| 7. References | 42 |
| Appendix I Patient Pill Calendar | |
| Appendix II Trametinib Ophthalmic Exam Form | 49 |
| Appendix III Actionable Mutations for Sub-Protocol EAY131-S2 | 51 |
| Appendix IV: Patient Clinical Trial Wallet Card | |

# TREATMENT SUBPROTOCOL CHAIR

Rev. Add25

Jason J. Luke, MD, FACP
University of Pittsburgh Medical Center and
Hillman Cancer Center
5150 Centre Ave. Room 563
Pittsburgh PA 15232
Phone: 412-623-4511

Fax: (412) 623-7948 E-mail: <u>lukejj@upmc.edu</u>

Rev.5/16

# TREATMENT SUBPROTOCOL CO-CHAIR

Hussein Abdul-Hassan Tawbi, MD, PhD
MD Anderson Cancer Center

Department of Melanoma Medical Oncology
1515 Holcombe Boulevard. Unit 0430
Houston, TX 77030
Phone: (713) 792-6111
Fax: (713) 745-1046
htawbi@mdanderson.org

# TRANSLATIONAL CHAIR

Andrew S. Chi, MD, PhD
Laura and Isaac Perlmutter Cancer Center
NYU Langone Medical Center
240 E. 38th Street, 19th Floor
New York, NY 10016
Phone: (646) 501-4802
Fax: (646) 754-9696

chia01@nyumc.org

# Schema



Cycle = 28 days Accrual Goal: 35

# EAY131-S2

Version Date: August 19, 2020

# 1. Introduction

# 1.1 <u>Trametinib Dimethyl Sulfoxide (GSK1120212B, MEKINIST)</u>

The RAF-MEK-ERK pathway plays a critical role in multiple cellular functions. Activation of the pathway can result from activation/mutations of the upstream receptor tyrosine kinases (RTKs) and RAS, or upregulation/mutations in RAF and MEK. Upon activation, RAF acts as the MAPK kinase kinase and activates MAPKK (MEK1/2), which in turn catalyze activation of the effectors ERK1/ERK2. Once activated, ERK1/2 translocate into the nucleus and phosphorylate a number of effector proteins and transcriptional factors that regulate cell proliferation, motility, differentiation, and survival.

Trametinib Dimethyl Sulfoxide (hereafter, referred to as trametinib) is one of the several MEK inhibitors in clinical development. On May 29, 2013, the U.S. Food and Drug Administration (FDA) approved trametinib for the treatment of patients with unresectable or metastatic melanoma with BRAF V600E or BRAF V600K mutations as detected by an FDA-approved test (U.S. Food and Drug Amdinistration, 2013). On January 10, 2014, the FDA granted accelerated approval to trametinib and dabrafenib for use in combination to treat patients with unresectable or metastatic melanoma with a BRAF V600E or V600K mutation as detected by an FDA-approved test (U.S. Food and Drug Administration, 2014).

Experience to date indicates that MEK is a valid target. In a phase 3 trial comparing trametinib with dacarbazine or paclitaxel in patients with BRAF V600E or V600K mutant metastatic melanoma, trametinib demonstrated a significantly better response rate, progression-free survival, and overall survival (Flaherty et al., 2012). Extensive research is underway to identify the patient selection markers and to develop rational combination strategies. Preclinical studies have provided strong rationale and proof of principle for combination of MEK inhibitors with RTK inhibitors (EGFR or IGF-1R) (Gopal et al., 2010; Ebi et al., 2011), PI3K/AKT inhibitors (Engelman et al., 2008; Hoeflich et al., 2009), and mTOR inhibitors. On the other hand, the optimal dose/schedule and patient selection criteria for combination regimens have not been defined. Phase 1 results for a number of combinations have been reported, including AZD6244 + MK2206 (Tolcher et al., 2011) and GDC-0973 + GDC-094 (MEK + PI3K inhibitor) (Bendell et al., 2011). In addition, efforts have focused on identifying other up stream mutations in cancers like GNAQ and GNA11, which may benefit from selective MEK inhibition.

# 1.1.1 Mechanisms of Action and Preclinical Data with Trametinib

Trametinib is a dimethyl sulfoxide (DMSO) solvate compound (ratio 1:1) with potent, allosteric and ATP non-competitive inhibition of MEK1/2 (IC50 of 0.7 and 0.9 nM against MEK1 and MEK2, respectively) (Gilmartin *et al.*, 2011). Trametinib inhibited MEK1/2 kinase activity and prevented RAF-dependent MEK phosphorylation (S217 for MEK1), producing prolonged pERK1/2 inhibition. Trametinib showed better potency against unphosphorylated MEK1/2 (u-MEK1/2) when compared with preactivated diphosphorylated MEK (pp-MEK), suggesting that u-MEK affords a higher affinity binding site for trametinib than does pp-MEK.

The specificity of trametinib was confirmed against a panel of 183 kinases, including MEK5 (the closet kinase homolog to MEK1/2), CRAF, BRAF, ERK1, and ERK2 (Yamaguchi *et al.*, 2011). Trametinib demonstrated equal potency against activated MEK1- and MEK2-mediated phosphorylation of ERK (sequence identity of 85% across the whole protein and 100% in the active site for humans). Trametinib demonstrated preferential inhibition of RAF-mediated MEK1 activation (IC $_{50}$  = 0.60 nM) over pMEK1 kinase activity (IC $_{50}$  = 13 nM) (Investigator's Brochure, 2012a).

BRAF-mutant Colo205, A375P F11s, and HT-29 human tumor xenograft mouse models showed the most significant mean tumor growth inhibition (TGI) (80% to 87%) at 3.0 mg/kg trametinib, with multiple complete and partial tumor regressions. In the Colo205 model, tumor regression was observed even at a dose of 0.3 mg/kg (Yamaguchi *et al.*, 2011). Two KRAS-mutant xenograft models, HCT-116 and A549, also showed significant TGI (83% and 75%) but without significant tumor regressions (Gilmartin *et al.*, 2011). As predicted by cell proliferation assays, tumor xenograft lines with wild-type (wt) RAF/RAS (PC3, BxPC3, and BT474) were much less sensitive, showing only modest TGI (44-46%) with no tumor regressions.

Pharmacodynamic studies were performed in mice treated with trametinib for 14 days (Gilmartin *et al.*, 2011). In the A375P F11s xenograft model, the first dose of trametinib (3 mg/kg) significantly reduced pERK for more than 8 hours on Day 1. pERK inhibition was more sustained (over 24 hours) after the Day 7 dose, probably due to an increase in the steady-state levels of trametinib after repeated doses. The average  $C_{\text{max}}$  in blood was 1,410 nM on Day 7, with an estimated half-life ( $t_{1/2}$ ) of 33 hours. In addition, immunohistochemistry (IHC) also confirmed inhibition of cell proliferation (reduced Ki67) and G1 cell cycle arrest (elevated p27Kip1/CDKN1B) following 4 days of treatment.

# 1.1.2 Clinical Pharmacokinetics (PK) and Activity of Trametinib

Phase 1 Trial of Trametinib Monotherapy (MEK111054)

There were 3 parts in this industry sponsored study. Part 1: The dose-escalation portion involved administration of trametinib (repeat doses of 0.125 mg to 4.0 mg) to patients with solid tumors or lymphoma in one of three schedules - (1) QD for 21 days followed by 7 days without drug, (2) loading dose on Day 1 or Day 1-2, followed by QD with the designated dose, or (3) QD dosing without a drug holiday. Part 2: cohort expansion at the recommended phase 2 dose (RP2D) for pancreatic cancer, melanoma, non-small cell lung cancer (NSCLC), colorectal cancer (CRC), or any BRAF mutation-positive cancer. Part 3: expansion to characterize the biologically active range of trametinib via analysis of pharmacodynamic biomarkers (biopsies or FDG-PET). The study has been completed and all parts, other than FDG-PET results, have been reported

The MTD of trametinib was established as 3 mg QD, but the recommended phase 2 dose (RP2D) was chosen at 2 mg QD based on tolerability of repeated cycles (Infante et al., 2012).

### PK and metabolism of trametinib:

PK measurements were conducted under fasting conditions. After a single dose (Day 1), AUC<sub>0-24</sub> and C<sub>max</sub> values were dose-proportional up to 6 mg, lower than dose proportional following 8 mg, and greater than dose proportional following the 10 mg dose. Median T<sub>max</sub> was 1.5 hours.

After repeat doses (Day 15), trametinib accumulated with a mean accumulation ratio of 6.6 at the RP2D of 2 mg QD. Between-subject variability in exposure ranged from 27-50% for C<sub>max</sub> and 20-41% for AUC<sub>0-24</sub> across all dosing regimens. The effective t<sub>1/2</sub> was approximately 4.5 days, and steady state was reached by approximately Day 15. Trametinib had a small peak:trough ratio of ~2 (Infante et al., 2010). At 2 mg QD on Day 15, mean AUC<sub>0-24</sub> was 376 ng•h/mL and C<sub>max</sub> 23 ng/mL, and the mean trough concentrations ranged from 10.0 to 18.9 ng/mL. The long half-life and small peak:trough ratio of trametinib allowed constant target inhibition within a narrow range of exposure.

# Drug-drug interactions:

Trametinib is metabolized predominantly via deacetylation (noncytochrome P450 [CYP450]-mediated) with secondary oxidation or in combination with glucuronidation biotransformation pathways (Investigator's Brochure, 2012a). The deacetylation is likely mediated by hydrolytic esterases, such as carboxylesterases, or amidases. Based on in vitro studies, trametinib is not an inhibitor of CYP1A2, CYP2A6, CYP2B6, CYP2D6, and CYP3A4. Trametinib dimethyl sulfoxide is a weak CYP2C8 inhibitor and weak CYP3A4 inducer. Drug-drug interactions with sensitive substrates of 2C8 and 3A4 are not anticipated. Trametinib has an overall low potential for drug-drug interactions.

# Pharmacodynamic effect and biomarkers:

The relationship between dose and tumor biomarkers such as pERK, Ki67, and p27, were evaluated in patients with BRAF or NRAS mutation-positive metastatic melanoma (Investigator's Brochure, 2012a). In general, increasing exposures and/or doses provided greater pharmacodynamic effects. The median change observed at a dose of 2 mg QD was 62% inhibition of pERK, 83% inhibition of Ki67, and a 175% increase in p27.

# Antitumor Activity in the phase 1 trial:

In the phase 1 trial, 14 patients with BRAF-mutant melanoma received trametinib at 2 mg QD. The overall objective response rate (ORR) was 43% (6/14), including 2 complete responses (CRs) (Investigator's Brochure, 2012a). In 9 patients with BRAF wt melanoma, 2 patients achieved a partial response (PR), and 3 stable disease (SD) (Infante et al., 2010). In 26 evaluable pancreatic cancer patients, there were 2 PRs (1 PR was KRAS mutation-positive) and 11 SD (2 achieved

EAY131-S2 Version Date: August 19, 2020

≥ 20% tumor reduction) (Messersmith et al., 2011). Among the 27 CRC patients (without selection of RAS or RAF mutations), 8 SD were observed.

# Antitumor Activity in Melanoma

Phase 3 trial of trametinib vs. chemotherapy in advanced V600 mutant melanoma:

In a phase 3 trial, patients with unresectable stage IIIC or IV cutaneous melanoma with a BRAF V600E or V600K mutation were randomized (2:1) to trametinib (2 mg, PO, QD) or chemotherapy (dacarbazine or paclitaxel) (Flaherty et al., 2012; MEKINIST, 2013). There were 322 patients in the intention-to-treat (ITT) population, of whom 273 (85%) were in the primary efficacy population (patients with BRAFV600E-positive cancer who did not have brain metastases at baseline). Of the patients, 214 were randomized to receive trametinib, and 108 were randomized to receive chemotherapy. Investigator-assessed efficacy data are summarized as follows:

| | Trametinib<br>(n=214) | Chemotherapy (DTIC)<br>(n=108) |
|---|---|---|
| PFS | | |
| Median, months (95% CI) | 4.8 (4.3, 4.9) | 1.5 (1.4, 2.7) |
| HR (95% CI) | 0.47 (0.34, 0.65) | |
| P value (log-rank test) | <i>P</i> < 0.0001 | |
| Confirmed Tumor Responses | | |
| Objective Response Rate (95% CI) | 22% (17, 28) | 8% (4, 15) |
| CR, n (%) | 4 (2%) | 0 |
| PR, n (%) | 43 (20%) | 9 (8%) |
| Duration of response | | |
| Median, months (95% CI) | 5.5 (4.1, 5.9) | NR (3.5, NR) |

CI = confidence interval; CR = complete response; HR = hazard ratio; NR = not reached; PFS = progression-free survival; PR = partial response

The 6-month OS rate was 81% in the trametinib group and 67% in the chemotherapy group. Mature data on OS are pending.

# <u>Experience with Trametinib in Metastatic Melanoma Following BRAF</u> Inhibitor Therapy

The clinical activity of single-agent trametinib was evaluated in a single-arm, multicenter, international trial in 40 patients with BRAF V600E or V600K mutation-positive, unresectable, or metastatic melanoma who had received prior treatment with a BRAF inhibitor. All patients received trametinib at a dose of 2 mg PO QD until disease progression or unacceptable toxicity. None of the patients achieved a confirmed PR or CR.

In a phase 1/2 monotherapy study, acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) patients were given trametinib at dose levels from 1-2 mg QD. Drug-related AEs in 45 patients were similar to that observed in patients with solid tumors, and 2 mg PO QD was selected for further investigation in this patient population. Twelve patients (23%) withdrew due to an AE, including cardiac failure (2) and infection (2). Efficacy was reported in 39 patients (Borthakur *et al.*, 2010). The best response in 13 patients with KRAS or NRAS mutations included 3 CRs (23%), 7 SD (54%), and 1 PD (progressive disease) (5%). In 26 patients with wild-type RAS or an unknown mutation, there were 2 PRs (8%).

In a multicenter phase 2 study, NSCLC patients with KRAS mutant tumors were randomized 2:1 to receive trametinib (2 mg QD) or docetaxel (75 mg/m² IV every 3 weeks) (Blumenschein *et al.*, 2013). A total of 134 pts were randomized to trametinib (89) or docetaxel (45); 129 patients had KRAS-mutant NSCLC. The hazard ratio for PFS was 1.14 (95% CI, 0.75-1.75; *P*=0.5197) with a median PFS of 11.7 versus 11.4 weeks for trametinib versus docetaxel. The overall response rate (ORR) was 12% for trametinib and 12% for docetaxel.

In a double-blind, phase 2 study evaluating the combination of gemcitabine with trametinib, untreated pancreatic cancer patients were randomized to receive gemcitabine (1000 mg/m² weekly  $\times$ 7 for 8 weeks, then weekly  $\times$ 3 every 4 weeks) plus either trametinib 2mg or placebo QD (Infante et al., 2013). Median OS was 8.4 months with trametinib compared to 6.7 months with placebo. Median PFS was 16 weeks versus 15 weeks, and ORRs and median duration of responses were 22% and 23.9 weeks and 18% and 16.1 weeks on trametinib and placebo; the median OS and ORR in the subgroup of patients with KRAS mutations (143/160) was similar to OS and ORR for all randomized patients.

The guanine nucleotide-binding protein G(q) subunit alpha (GNAQ) and guanine nucleotide-binding protein subunit alpha-11 (GNA11) are large GTPases of the Gqq family (Van Raamsdonk et al., 2009; Van Raamsdonk et al., 2010). Recurrent activating mutations in GNAQ (3.3% of 8778 cancer samples in COSMIC v63) or GNA11 (2.3% OF 6237 cancers in COSMIC v62) have been identified in cancers. Most of these mutations result in defective GTPase activity and render the proteins constitutively active (O'Hayre et al., 2013). Activating mutations ultimately lead to downstream activation of MAPK signaling (Hubbard and Hepler, 2006; Griner and Kazanietz, 2007). The highest prevalence of GNAQ and GNA11 mutations are found in uveal melanoma (33% AND 39% respectively), blue nevi (32% and 3-5%, respectively) and cutaneous melanoma (1.4% and 1.3%, respectively), but are also found in colon adenocarcinoma at about 2%.(Shoushtari AN et al GNAQ and GNA11 mutations in uveal melanoma. Melanoma Res 2014; 24: 525-534). MEK inhibitors can be active in melanomas with GNAQ or GNA11 mutations. Preclinical activity of the MEK 1 and 2 inhibitor selumetinib has been published

(Ambrosini et al. Identification of unique MEK dependent genes in GNAQ mutant uveal melanoma involved in cell growth, tumor cell invasion and MEK resistance. Clin Cancer Res 2012; 18: 3552-3561). A subsequent randomized phase II trial of investigator's choice chemotherapy with or without selumetinib in metastatic uveal melanoma showed, in an unplanned analysis, a significant improvement in PFS for the selumetinib group (Carvajal RD, Sosman JA, Quevedo JF, Milhem MM, Joshua AM,

Kudchadkar RR, et al. Effect of selumetinib vs chemotherapy on progressionfree survival in uveal melanoma: a randomized clinical trial. JAMA 2014; 311:2397–2405). In a phase I study of trametinib in patients with melanoma, combined exploratory and clinical genotyping of patients who entered the trial with uveal melanoma revealed 6 patients with GNAQ or GNA11 mutations. 50% had response of stable disease and one patient with a GNA11 mutation remained on trametinib for more than 40 weeks (Falchook GS et al. Activity of the oral MEK inhibitor trametinib in patients with advanced melanoma: a phase 1 dose escalation trial. Lancet Oncol 2012; 13: 782-89).

# 1.2 Supporting Preliminary Data

# **GNAQ / GNA11** Biology and Targeted Therapy

The guanine nucleotide-binding protein G(q) subunit alpha (GNAQ) and guanine nucleotide-binding protein subunit alpha-11 (GNA11) are two closely related large GTPases of the Gαg family (Van Raamsdonk et al., 2009; Van Raamsdonk et al., 2010). Mutations in GNAQ or GNA11 are likely to be present in 1.6 - 2% of the population of cancer patients based on the cBIO Portal database. Mutations in *GNAQ* or *GNA11* eliminate the activity of the heterotrimeric G protein α subunits Gag and Gall GTPase, leading to hyperactivation of signaling downstream of the GNAQ and GNA11 (O'Hayre et al., 2013). The oncogenic activity of GNAQ was initially revealed as part of a systematic analysis of the transforming potential of G proteins and their coupled receptors (Kalinec et al., 1992). The best-described signaling event downstream of Gαg involves activation of phospholipase C (PLC) with subsequent increase in inositol 1,4,5trisphosphate (IP3), and diacylglycerol (DAG) (Hubbard and Hepler, 2006). IP3 increases cytoplasmic Ca2+ levels leading to modulation of multiple calciumregulated pathways. Together with DAG, this stimulates classical protein kinase C (PKC) isoforms (Griner and Kazanietz, 2007). GNAQ thus utilizes PLC to stimulate MAPK.

Based upon the finding that uveal melanoma (UM) is characterized by functionally active mutations in GNAQ or GNA11 (Ivey et al., 2003; Onken et al., 2008; Raamsdonk et al., 2008), as well as preclinical findings demonstrating antitumor effects of MEK inhibition in *GNAQ/GNA11* mutant UM (Ambrosini et al., 2012), a randomized trial of the MEK inhibitor selumetinib versus temozolomide was performed in patients with UM. The primary endpoint of the study, progression-free survival, was doubled as compared with chemotherapy. A hazard ratio for progression of 0.46 in favor of selumetinib was observed (Carvajal et al., 2013). The overall response for patients whose tumors harbored *GNAQ/GNA11* mutations was 15%. The overall response rate was zero in patients who crossed over to selumatinib after failure of temozolomide. Patients experiencing RECIST responses and tumor shrinkage form baseline were found

to harbor mutations in the Q209L; Q209P; Q209H; and Q209R of exon 5 as well as R183 of exon 4 of *GNAQ* (personal communication from Richard Carvajal, MD)

The preliminary success of the MEK inhibitor selumetinib in targeting GNAQ/GNA11 suggests that MAPK inhibition is a reasonable therapeutic target in UM and other GNAQ/11 mutant cancers. Two approaches may be considered in improving the clinical outcome of patients then including adding a second signaling inhibitor to a MEK inhibitor or alternatively, more completely suppressing MAPK signaling with a more potent MEK inhibitor. In considering combination approaches, it is important to make note that signaling downstream of GNAQ/GNA11 is mediated through PKC isoforms, this molecule has been of interest for targeted therapy development in this molecular model. Inhibitors of PKC such as sotrastaurin and related compounds, selectively block the proliferation of melanoma cell lines with mutations in GNAQ or GNA11 (Wu et al., 2012a; Wu et al., 2012c). Similar results are observed with human melanoma cell lines with GNAQ or GNA11 mutations. While MEK inhibitors suppress the growth of UM cell lines, they show no selectivity compared to melanoma cell lines with mutations in other oncogenes such as RAS or BRAF. By contrast, in UM with GNAQ or GNA11 mutations, a combination of PKC inhibition and MEK inhibitors leads to a highly synergistic effect. These results suggest that combined inhibition of PKC and MEK may represent a rational combination to be evaluated in GNAQ and GNA11 mutant cancers.

Combination approaches of MEK inhibition with other pathway inhibitors have also been examined in *GNAQ* or *GNA11* mutant uveal melanoma. Based upon preclinical data demonstrating enhancement of MEK inhibitor-induced antitumor effects by concurrent inhibition of AKT or PI3K (Ambrosini et al., 2013; Khalili et al., 2012), a phase II trial of trametinib in combination with GSK2141795, an oral AKT inhibitor, was launched (NCI 9445). Furthermore, building upon preclinical data demonstrating the enhanced susceptibility of tumor cells to chemotherapy with concurrent MEK inhibition (Holt et al., 2012), as well as the greater PFS observed with the combination in a study of cutaneous melanoma (Holt et al., 2012; Robert et al., 2013), a phase II trial of DTIC with or without selumetinib has also begun accrual (NCT01974752).

To date, combination approaches of molecular inhibitors have proved to be toxic relative to expectations for targeted therapies (Bendell et al., 2014). Therefore, consideration of MAPK suppression by a higher potency MEK inhibitor would be reasonable. As above, selumetinib demonstrated a clinically significant response rate of 15% in UM. Selumetinib in a MEK1/2 inhibitor with MEK1 IC 50 of 10 ηM. Other MEK inhibitors are available including the MEK1/2 inhibitor trametinib. which demonstrates a MEK1 IC<sub>50</sub> of 0.7 ηM (Luke et al. 2014). Trametinib has not been evaluated in UM or GNAQ/11 mutant tumors in a robust manner. In the single agent phase I study of trametinib (Infante et al., 2012), 16 patients with UM were treated without identification of any partial response. However, the GNAQ/11 mutational status of these patients was not disclosed. Whereas in the selumetinib phase II trial, patients were untreated, in the trametinib phase I study the median number of prior therapies was 3. This likely impacted on the result. Of the 16 patients treated, best response included 8 patients with stable disease with 4 patients on treatment greater than 16 weeks. This decrease in efficacy of MEK inhibition after further lines of therapy is consistent with what was seen in the selumetinib trial. In that study, no patients who received chemotherapy first

had a response to selumetinib after crossing over on the study. The molecular mechanism underpinning this change in biology is unknown though it has been postulated that perhaps the essential signaling pathways in UM can change after chemotherapy. An on-going study is evaluating trametinib with and without an AKT inhibitor in untreated advanced UM. This prior experience with MEK inhibitors suggests that treatment with trametinib for UM and *GNAQ/11* mutant tumors may be efficacious and is an important clinical question to explore. Trametinib is chosen for this study in place of selumatinib because of its better efficacy based on cross trial comparison for similar patient population (BRAFV600E melanoma).

# EAY131-S2

Version Date: August 19, 2020

# 2. Selection of Patients

Each of the criteria in the checklist that follows must be met, along with the eligibility in the main screening study, in order for a patient to be considered eligible for this study. Use the checklist to confirm a patient's eligibility. For each patient, this checklist must be photocopied, completed and maintained in the patient's chart.

In calculating days of tests and measurements, the day a test or measurement is done is considered Day 0. Therefore, if a test is done on a Monday, the Monday four weeks later would be considered Day 28.

| | ECOG-AC | CRIN Patient No. |
|---|---|---|
| | | nitials (L, F, M) |
| | | Signature and Date |
| | NOTE: | All CTEP Policy does not allow for the issuance of waivers to any protocol specified criteria ( <a href="http://ctep.cancer.gov/protocolDevelopment/policies_deviations.htm">http://ctep.cancer.gov/protocolDevelopment/policies_deviations.htm</a> ). Therefore, all eligibility criteria listed in Section 2 must be met, without exception. The registration of individuals who do not meet all criteria listed in Section 2 can result in the participant being censored from the analysis of the study, and the citation of a major protocol violation during an audit. All questions regarding clarification of eligibility criteria must be directed to the Group's Executive Officer ( <a href="EA.Execofficer@jimmy.harvard.edu">EA.Execofficer@jimmy.harvard.edu</a> ) or the Group's Regulatory Officer ( <a href="EA.Execofficer@jimmy.harvard.edu">EA.RegOfficer@jimmy.harvard.edu</a> ). |
| | NOTE: | Institutions may use the eligibility checklist as source documentation if it has been reviewed, signed, and dated prior to registration/randomization by the treating physician. |
| | NOTE: | All patients must have signed the relevant treatment consent form |
| | 2.1 <u>Elig</u> | gibility Criteria: |
| | 2.1 | Patients must fulfill all eligibility criteria outlined in Section 3.1 of MATCH Master Protocol (excluding Section 3.1.6) at the time of registration to treatment step (Step 1, 3, 5, 7). |
| Rev. Add13 | 2.1 | 1.2 Patients must have GNAQ or GNA11 mutations, or another aberration, as determined via the MATCH Master Protocol and according to Appendix III. See <a href="Appendix III">Appendix III</a> for information on the targeted mutations and corresponding Levels of Evidence. |
| | 2.1 | <ul> <li>Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:</li> <li>Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block).</li> <li>Treatment-refractory hypertension defined as a blood pressure of systolic &gt; 140 mmHg and/or diastolic &gt;90 mmHg which cannot be controlled by anti-hypertensive therapy.</li> </ul> Date of ECG: |
| Rev. Add13 | 2.1 <u>Eliq</u> 2.1 | All patients must have signed the relevant treatment consent form gibility Criteria: 1.1 Patients must fulfill all eligibility criteria outlined in Section 3.1 of MATCH Master Protocol (excluding Section 3.1.6) at the time of registration to treatment step (Step 1, 3, 5, 7). 1.2 Patients must have GNAQ or GNA11 mutations, or another aberration, as determined via the MATCH Master Protocol and according to Appendix III. See Appendix III for information on the targeted mutations and corresponding Levels of Evidence. 1.3 Patients must have an electrocardiogram (ECG) within 8 weeks proto treatment assignment and must have NONE of the following cardiac criteria: • Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block). • Treatment-refractory hypertension defined as a blood pressure systolic > 140 mmHg and/or diastolic >90 mmHg which cannot controlled by anti-hypertensive therapy. |

**OPTIONAL:** This signature line is provided for use by institutions wishing to use the eligibility checklist as source documentation.

# 3. Treatment Plan

# 3.1 Administration Schedule

All patients will receive trametinib 2mg daily continuously until intolerable toxicity, disease progression, or the end of the study.

Trametinib should be administered once per day, continuously; and should be taken at about the same time each day. The study drug should be administered together with approximately eight ounces of water. Trametinib should be taken fasting, at least 1 hour before or 2 hours after a meal. If a subject vomits after taking study medication, the subject should be instructed not to retake the dose and should take the next scheduled dose.

If a dose of trametinib is missed, only take the dose if it is more than 12 hours until the next scheduled dose.

Trametinib should be stored at 2-8°C (36-46°F). Refrigerate. Do not freeze.

# 3.2 Adverse Event Reporting Requirements

The Adverse Event Reporting Requirements for all EAY131 subprotocols are outlined in the MATCH MASTER protocol. Please refer to those guidelines when determining if an event qualifies as a Serious Adverse Event (SAE) and requires expedited reporting via CTEP's Adverse Event Reporting System (CTEP-AERS).

In addition, the following section outlines agent specific requirements and must be followed to ensure all reporting requirements are met.

3.2.1 Additional instructions, requirements and exceptions for protocol EAY131-Subprotocol S2.

# **Additional Instructions**

For instructions on how to specifically report events that result in persistent or significant disability/incapacity, congenital anomaly, or birth defect events via CTEP-AERS, please contact the AEMD Help Desk at <a href="mailto:aemd@tech-res.com">aemd@tech-res.com</a> or 301-897-7497. This will need to be discussed on a case-by-case basis.

# EAY131- Subprotocol S2 specific expedited reporting requirements:

- LVEF Changes: If any of the following circumstances occur, the event(s) must be reported via CTEP-AERS according to the timeframes outlined in the AE table in section 5.3.6 of the MATCH Master protocol
  - Asymptomatic: Absolute decrease of >10% in LVEF compared to baseline and ejection fraction below the institution's LLN and LVEF does not recover within 4 weeks
  - Symptomatic: Grade 3-4 LVEF

Rev. 12/16

Please refer to the dose modification instructions for further information regarding Treatment Modification and Management Guidelines for LVEF Decrease

- Visual Changes: If RPED (retinal pigment epithelial detachments) or RVO (retinal vein occlusion) are diagnosed, the event(s) must be reported via CTEP-AERS according to the timeframes outlined in the AE table in section 5.3.6 of the MATCH Master protocol. Please refer to the dose modification instructions for further information regarding Treatment Modification and Management Guidelines for Visual Changes.
- Liver Chemistry Changes: If any of the following circumstances occur, the event(s) must be reported via CTEP-AERS according to the timeframes outlined in the AE table in section 5.3.6 of the MATCH Master protocol
  - ALT ≥ 3xULN and bilirubin ≥ 2x ULN or > 35% direct bilirubin
  - ALT ≥ 3xULN and INR ≥ 1.5, if INR measured (INR threshold does not apply if subject is on anticoagulant)
- Please refer to the dose modification instructions for further information regarding Treatment Modification and Management Guidelines for Liver Chemistry Changes
- Pregnancies: Pregnancies and suspected pregnancies (including a positive or inconclusive pregnancy test, regardless of age or disease state) occurring while the female patient is on Trametinib, or within 28 days of the patient subject's last dose of Trametinib, are considered immediately reportable events. The pregnancy, suspected pregnancy, or positive/ inconclusive pregnancy test must be reported via CTEP-AERS within 24 hours of the Investigator's knowledge. Please refer to Appendix VIII in MATCH Master protocol for detailed instructions on how to report the occurrence of a pregnancy as well as the outcome of all pregnancies.

# EAY131-S2 specific expedited reporting exceptions:

For study Subprotocol S2, the adverse events listed below **do not** require expedited reporting via CTEP-AERS:

- If an AE meets the reporting requirements of the protocol, and it is listed on the SPEER, it should <u>ONLY</u> be reported via <u>CTEP-AERS</u> if the grade being reported exceeds the grade listed in the parentheses next to the event
- 3.2.2 Second Primary Cancer Reporting Requirements

NOTE: The MATCH Master Protocol outlines the standard requirements for the reporting of second primaries. Please be aware that there are additional requirements for this subprotocol. Please adhere to the guidelines outlined below for the reporting of second primaries on this subprotocol.

Rev. 5/16

Rev. Add25

All cases of second (second malignancy is a cancer that is unrelated to any prior anti-cancer treatment, including the treatment on this protocol) **and** secondary malignancies (secondary malignancy is a cancer caused by any prior anti-cancer treatment, including the treatment on this protocol), including acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS)], regardless of attribution, that occur following treatment on NCI-sponsored trials must be reported as follows:

- 1. Complete a Second Primary Form in Medidata Rave within 14 days.
- 2. Report the diagnosis via CTEP-AERS, regardless of attribution, at <a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>

Report under a.) leukemia secondary to oncology chemotherapy, b.) myelodysplastic syndrome, or c.) treatment related secondary malignancy

- 3. Upload a copy of the pathology report to ECOG-ACRIN via Medidata Rave and submit a copy to NCI/CTEP confirming the diagnosis.
- If the patient has been diagnosed with AML/MDS, upload a copy of the cytogenetics report (if available) to ECOG-ACRIN via Medidata Rave and submit a copy to NCI/CTEP.

NOTE: All new malignant tumors must be reported through CTEP-AERS whether or not they are thought to be related to either previous or current treatment. All new malignancies should be reported including solid tumors (including non-melanoma skin malignancies), hematologic malignancies, Myelodysplastic Syndrome (MDS)/Acute Myelogenous Leukemia (AML), and in situ tumors.

Whenever possible, the CTEP-AERS report should include the following:

- tumor pathology
- history of prior tumors
- prior treatment/current treatment including duration
- any associated risk factors or evidence regarding how long the tumor may have been present
- when and how the tumor was detected
- molecular characterization or cytogenetics or the original tumor (if available) and of any new tumor
- tumor treatment and outcome (if available)

**NOTE:** The Second Primary Form and the CTEP-AERS report should not be used to report recurrence or development of metastatic disease.

NOTE: If a patient has been enrolled in more than one NCIsponsored study, the Second Primary Form must be submitted for the most recent trial. ECOG-ACRIN must be provided with a copy of the form and the associated

pathology report and cytogenetics report (if available) even if ECOG-ACRIN was not the patient's most recent trial.

NOTE:

Once data regarding survival and remission status are no longer required by the protocol, no follow-up data should be submitted via CTEP-AERS or by the Second Primary Form.

Rev. 1/17 Rev. Add19 Rev. Add25

# 3.3 Comprehensive Adverse Events and Potential Risks List (CAEPR) for Trametinib dimethyl sulfoxide (GSK1120212B, NSC 763093)

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements' <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/docs/aeguidelines.pdf</a> for further clarification. *Frequency is provided based on 1111 patients*. Below is the CAEPR for Trametinib dimethyl sulfoxide (GSK1120212B).

NOTE:

If an AE meets the reporting requirements of the protocol, and it is listed on the SPEER, it should **ONLY** be reported via CTEP-AERS if the grade being reported exceeds the grade listed in the parentheses next to the event.

Version 2.6, October 10, 20191

| Relat | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| | Less Likely (<=20%) PHATIC SYSTEM DISORD | Rare but Serious (<3%) | |
| BLOOD AND LYWP | | JERS<br>I | 4 |
| 04 0014 0 010 000 | Anemia | | Anemia (Gr 3) |
| CARDIAC DISORDI | ERS | T., | |
| | | Heart failure | |
| | | Left ventricular systolic | |
| | | dysfunction | |
| | Sinus bradycardia | | |
| EYE DISORDERS | | | |
| | Blurred vision | | |
| | Dry eye | | |
| | | Eye disorders - Other<br>(chorioretinopathy also<br>known as retinal pigment<br>epithelial detachment) | |
| | | Eye disorders - Other (retinal vein occlusion) | |
| | Eye disorders - Other (visual disorders) <sup>2</sup> | | |
| | | Papilledema | |
| | Periorbital edema | | |
| <b>GASTROINTESTINA</b> | AL DISORDERS | | |
| | Abdominal pain | | Abdominal pain (Gr 2) |
| | | Colitis | |
| | | Colonic perforation | |
| | Constipation | · | Constipation (Gr 2) |

| Relat | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| Diarrhea | | | Diarrhea (Gr 3) |
| | Dry mouth | | Dry mouth (Gr 2) |
| | Dyspepsia | | Dyspepsia (Gr 2) |
| | Mucositis oral | | Mucositis oral (Gr 3) |
| Nausea | | | Nausea (Gr 3) |
| | Vomiting | | Vomiting (Gr 3) |
| GENERAL DISORD | ERS AND ADMINISTRAT | ION SITE CONDITIONS | |
| | Chills | | Chills (Gr 2) |
| | Edema face | | |
| Fatigue | | | Fatigue (Gr 3) |
| | Fever | | Fever (Gr 2) |
| Generalized edema | | | Generalized edema <sup>3</sup> (Gr 2) |
| IMMUNE SYSTEM | | | |
| | Allergic reaction <sup>4</sup> | | |
| INFECTIONS AND I | | | |
| | Folliculitis | | Folliculitis (Gr 2) |
| | Lung infection | | |
| | Paronychia | | Paronychia (Gr 2) |
| | Skin infection | | Skin infection (Gr 2) |
| INVESTIGATIONS | | | |
| | Alanine<br>aminotransferase<br>increased | | Alanine aminotransferase increased (Gr 3) |
| | Alkaline phosphatase increased | | Alkaline phosphatase increased (Gr 2) |
| | Aspartate<br>aminotransferase<br>increased | | Aspartate<br>aminotransferase<br>increased (Gr 3) |
| | CPK increased Ejection fraction decreased | | |
| METABOLISM AND | NUTRITION DISORDER | S | |
| WE IT ESCIONITAINE | Anorexia | T | Anorexia (Gr 3) |
| | Dehydration | | Dehydration (Gr 3) |
| | Hypoalbuminemia | | |
| | Hypomagnesemia | | Hypomagnesemia (Gr 2) |
| | Hyponatremia | | Hyponatremia (Gr 3) |
| MUSCULOSKELET | AL AND CONNECTIVE TI | SSLIE DISORDERS | nyponduenna (Or 3) |
| MOOODLOGKELL | Arthralgia | | |
| | Back pain | | Back pain (Gr 2) |
| | Pain in extremity | | Pain in extremity (Gr 2) |
| | i animiexuemilly | Rhabdomyolysis | rani in extremity (Gr 2) |
| NERVOUS SYSTEM | A DISODDEDS | T T I AD U O I I I J O I | |
| NEINVOUSSISIE | 1 | T | Dizzinogo (Cr 2) |
| | Dizziness | | Dizziness (Gr 2) |
| | Headache | | Headache (Gr 2) |

| Relat | Specific Protocol<br>Exceptions to Expedited<br>Reporting (SPEER) | | |
|---|---|---|---|
| Likely (>20%) Less Likely (<=20%) Rare but Serious (<3%) | | | |
| RESPIRATORY, TH | IORACIC AND MEDIASTI | NAL DISORDERS | |
| | Cough | | Cough (Gr 2) |
| | Dyspnea | | Dyspnea (Gr 3) |
| | | Pneumonitis | |
| SKIN AND SUBCUT | TANEOUS TISSUE DISOF | RDERS | |
| | Alopecia | | Alopecia (Gr 2) |
| | Dry skin | | Dry skin (Gr 2) |
| | Nail changes | | |
| | | Palmar-plantar<br>erythrodysesthesia<br>syndrome | |
| Pruritus | | Pruritus (Gr 2) | |
| | | Skin and subcutaneous<br>tissue disorders - Other<br>(drug reaction with<br>eosinophilia and systemic<br>symptoms [DRESS]) | |
| Skin and<br>subcutaneous<br>tissue disorders -<br>Other (rash) <sup>5</sup> | | | Skin and subcutaneous<br>tissue disorders - Other<br>(rash) <sup>5</sup> (Gr 3) |
| | | Stevens-Johnson<br>syndrome <sup>6</sup> | |
| VASCULAR DISOR | DERS | | |
| | Hypertension | | Hypertension (Gr 3) |
| | | Thromboembolic event (venous) | |
| | Vascular disorders -<br>Other (hemorrhage) <sup>7</sup> | | |

<sup>&</sup>lt;sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting PIO@CTEP.NCI.NIH.GOV. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>&</sup>lt;sup>2</sup>Visual disorders include visual disturbance that can be associated with conjunctival hemorrhage, corneal graft rejection, cyclitis, eye nevus, halo vision, iritis, macular edema, retinal hemorrhage, visual acuity reduced, visual impairment, and vitreous detachment.

<sup>&</sup>lt;sup>3</sup>Generalized edema includes edema, lymphedema, and edema limbs.

<sup>&</sup>lt;sup>4</sup>Hypersensitivity (allergic reactions) may present with symptoms such as fever, rash, increased liver function tests, and visual disturbances.

<sup>&</sup>lt;sup>5</sup>Skin and subcutaneous tissue disorders - Other (rash) may include rash, rosacea, rash acneiform, erythematous rash, genital rash, rash macular, exfoliative rash, rash generalized, erythema, rash papular, seborrhoeic dermatitis, dermatitis psoriasiform, rash follicular, skin fissures, and skin chapped.

<sup>&</sup>lt;sup>6</sup>Stevens-Johnson syndrome has been observed in patients treated with trametinib and dabrafenib combination.

EAY131-S2

Adverse events reported on trametinib dimethyl sulfoxide (GSK1120212B) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that trametinib dimethyl sulfoxide (GSK1120212B) caused the adverse event:

**BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Disseminated intravascular coagulation; Febrile neutropenia; Leukocytosis

CARDIAC DISORDERS - Atrial fibrillation: Cardiac arrest: Myocardial infarction: Restrictive cardiomyopathy; Sinus tachycardia

**EYE DISORDERS** - Corneal ulcer; Eyelid function disorder; Flashing lights; Floaters; Glaucoma; Photophobia

GASTROINTESTINAL DISORDERS - Ascites; Duodenal ulcer; Esophageal necrosis; Esophageal ulcer; Esophagitis; Gastric hemorrhage<sup>7</sup>; Gastric ulcer; Gastritis; Gastrointestinal disorders - Other (intestinal obstruction): Gastrointestinal disorders -Other (pneumatosis intestinalis): Gastrointestinal fistula: Gingival pain: Hemorrhoidal hemorrhage<sup>7</sup>; Ileus; Obstruction gastric; Pancreatitis; Small intestinal obstruction

**GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Flu like** symptoms; General disorders and administration site conditions - Other (axillary pain); Localized edema; Malaise; Non-cardiac chest pain; Pain

HEPATOBILIARY DISORDERS - Cholecystitis; Hepatic failure; Hepatic pain; Hepatobiliary disorders - Other (hepatic encephalopathy)

**INFECTIONS AND INFESTATIONS** - Biliary tract infection; Catheter related infection; Device related infection: Endocarditis infective: Enterocolitis infectious: Hepatitis viral: Infections and infestations - Other (abscess limb); Infections and infestations - Other (necrotizing fasciitis); Infections and infestations - Other (oral infection); Pharyngitis; Sepsis; Upper respiratory infection; Urinary tract infection

# INJURY, POISONING AND PROCEDURAL COMPLICATIONS - Bruising

**INVESTIGATIONS** - Blood bilirubin increased: Blood lactate dehydrogenase increased: Creatinine increased; Electrocardiogram QT corrected interval prolonged; GGT increased; Lipase increased; Lymphocyte count decreased; Platelet count decreased; Serum amylase increased; White blood cell decreased

METABOLISM AND NUTRITION DISORDERS - Hyperglycemia; Hyperkalemia; Hyperphosphatemia; Hyperuricemia; Hypocalcemia; Hypoglycemia; Hypokalemia

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Generalized muscle weakness; Muscle cramp; Musculoskeletal and connective tissue disorder - Other (compression fracture); Myalgia; Neck pain

NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND **POLYPS)** - Tumor hemorrhage<sup>7</sup>; Tumor pain

NERVOUS SYSTEM DISORDERS - Dysgeusia: Encephalopathy: Intracranial hemorrhage<sup>7</sup>; Lethargy; Nervous system disorders - Other (diplopia); Seizure; Somnolence; Stroke; Syncope; Transient ischemic attacks

**PSYCHIATRIC DISORDERS** - Anxiety; Confusion; Delirium; Depression; Hallucinations; Insomnia; Personality change

RENAL AND URINARY DISORDERS - Acute kidney injury; Cystitis noninfective; Dysuria; Hematuria; Proteinuria; Urinary incontinence

<sup>&</sup>lt;sup>7</sup>The majority of hemorrhage events were mild. Major events, defined as symptomatic bleeding in a critical area or organ (e.g., eye, GI hemorrhage, GU hemorrhage, respiratory hemorrhage), and fatal intracranial hemorrhages have been reported.

**REPRODUCTIVE SYSTEM AND BREAST DISORDERS** - Vaginal fistula; Vaginal hemorrhage<sup>7</sup>

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Bronchopulmonary hemorrhage<sup>7</sup>; Hypoxia; Laryngeal edema; Oropharyngeal pain; Pleural effusion; Pneumothorax; Productive cough; Pulmonary hypertension; Respiratory failure; Sinus disorder

**SKIN AND SUBCUTANEOUS TISSUE DISORDERS** - Bullous dermatitis; Photosensitivity; Purpura; Skin and subcutaneous tissue disorders - Other (erythema nodosum); Skin ulceration; Urticaria

VASCULAR DISORDERS - Hematoma; Hot flashes; Hypotension

**NOTE**: Trametinib (GSK1120212B) in combination with other agents could cause an exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either agent.

#### Rev. 12/16 3.4 **Dose Modifications**

NOTE: Patients who interrupt trametinib for > 2 weeks will be removed from this subprotocol, unless the interruption was for reduction in LVEF, visual changes or RPED with subsequent recovery as described in corresponding tables below.

All toxicity grades below are described using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP website (http://ctep.cancer.gov).

341 Dose Modification Guidelines for Trametinib Adverse Events of Special Interest

The dose levels for this study are provided in Table 1.

| Dose Levels | Trametinib once daily |
|--------------------------------|-----------------------|
| Full dose | 2 mg |
| 1st Dose reduction | 1.5 mg |
| 2 <sup>nd</sup> Dose reduction | 1.0 mg |

#### Table 1 **Dose Level Reduction Guidelines**

- 3.4.2 If an AE resolves to grade 1 or lower (or baseline) and remains grade 1 or lower at the reduced dose level and the subject does not experience any additional AEs requiring dose hold or reductions, then after 4 weeks of the study treatment at reduced dose, the dose of trametinib may be increased one dose level. If a dose reduction below 1 mg once daily for trametinib is required, then trametinib will be permanently discontinued.
- Guidelines for Cardiovascular Adverse Events 3.4.3

Cardiovascular adverse events have been seen in subjects receiving trametinib[4]). Guidelines for LVEF decreases and hypertension are provided below.

3.4.3.1 Left Ventricular Ejection Fraction (LVEF)

> Decreases of the left-ventricular-ejection-fraction (LVEF) have been observed in subjects receiving trametinib. Therefore, ECHOs (preferred) or MUGA's must be performed to assess cardiac ejection fraction. The procedure performed at baseline must be performed at all designated visits as outlined in the Time and Events Table (See Section 4.1).

> Dose modification guidance and stopping criteria for LVEF decrease are provided (Table 2).

Table 2 Dose Modification Guidelines and Stopping Criteria for LVEF Decrease

| | Clinic | LVEF-drop (%) or<br>CTCAE grade | Action and Dose Modification |
|---|---|---|---|
| | Asymptomatic | Absolute decrease of >10% in LVEF compared to baseline and ejection fraction below the institution's LLN | <ul> <li>Interrupt trametinib and repeat ECHO/MUGA within 2 weeks<sup>a</sup></li> <li>If the LVEF recovers within 4 weeks (defined as LVEF ≥ LLN and absolute decrease ≤ 10% compared to baseline): <ul> <li>Consult with the subprotocol Study Chair and request approval for restart</li> <li>Restart treatment with trametinib at reduced dose by one dose level<sup>b</sup></li> <li>Repeat ECHO/MUGA 2, 4, 8 and 12 weeks after re-start; continue in intervals of 12 weeks thereafter</li> </ul> </li> <li>If LVEF does not recover within 4 weeks <ul> <li>Consult with cardiologist</li> <li>Permanently discontinue trametinib</li> <li>Repeat ECHO/MUGA after 2, 4, 8, 12, and 16 weeks or until resolution</li> <li>Consult with the subprotocol Study Chair.<sup>c</sup></li> </ul> </li> </ul> |
| Rev. Add13 | Symptomatic <sup>b</sup> | Grade 3: resting LVEF<br>39-20% or > 20%<br>absolute reduction from<br>baseline<br>Grade 4: resting LVEF<br>< 20% | <ul> <li>Permanently discontinue trametinib.</li> <li>Report as SAE</li> <li>Consult with cardiologist</li> <li>Repeat ECHO/MUGA after 2, 4, 8, 12, and 16 weeks or until resolution</li> </ul> |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; ECHO = echocardiogram; GSK = GlaxoSmithKline; LLN = lower limit of normal; LVEF = left ventricular ejection fraction; MUGA=Multi-gated acquisition

- a. If ECHO/MUGA does not show LVEF recovery after 2 weeks, repeat ECHO/MUGA 2 weeks later.
- b. Escalation of trametinib to previous dose level can be considered if LVEF remains stable for 4 weeks after restarting of trametinib. Approval from the subprotocol Study Chair is required.
- c. Symptoms may include: dyspnea, orthopnea, and other signs and symptoms of pulmonary congestion and edema.

# 3.4.3.2 **Hypertension**

Increases in blood pressure (BP) have been observed in patients receiving trametinib. Recommendations for BP monitoring and management are provided below.

*Monitoring:* All BP assessments should be performed under the following optimal conditions:

- The subject has been seated with back support, ensuring that legs are uncrossed and flat on the floor
- The subject is relaxed comfortably for at least 5 minutes

- Restrictive clothing has been removed from the cuff area and the appropriate right size has been selected
- The subject's arm is supported so that the middle of the cuff is at heart level
- The subject remains quiet during the measurement.
- In subjects with an initial BP reading within the hypertensive range, a second reading should be taken at least 1 minute later, with the two readings averaged to obtain a final BP measurement. The averaged value should be recorded in the eCRF.
- Persistent hypertension is defined as an increase of systolic blood pressure (SBP) > 140 mm Hg and/or diastolic blood pressure (DBP) > 90 mm Hg in three consecutive visits with blood pressure assessments from two readings as described above. Visits to monitor increased blood pressure can be scheduled independently from the per-protocol visits outlined in the study calendar. Ideally, subsequent blood pressure assessments should be performed within one week.

Table 3 Management and Dose Modification Guidelines for Hypertension

| Management and Trametinib Dose Modification for Hypertension | |
|---|---|
| Event Management Guideline Do | Dose Modification |
| Definitions used in the table: | |

- <u>Persistent hypertension</u>: Hypertension detected in two separate readings during up to three subsequent visits.
- <u>Well-controlled hypertension:</u> Blood pressure of SBP ≤140 mmHg and DBP ≤90 mmHg in two separate readings during up to three subsequent visits.
- <u>Symptomatic hypertension</u>: Hypertension associated with symptoms (*e.g.*, headache, lightheadedness, vertigo, tinnitus, episodes of fainting or other symptoms indicative of hypertension) that resolve after the blood pressure is controlled within the normal range.

#### - Asymptomatic hypertension: SBP > 140 mmHg and/or DBP > 90 mmHg in the absence of the above symptoms. Continue trametinib at the current (Scenario A) Adjust current or initiate new antihypertensive medication(s). dose. Asymptomatic and persistent SBP of ≥ 140 and < 160 mmHg. Titrate antihypertensive or DBP ≥ 90 and < 100 mmHg, medication(s) during the next 2 weeks to achieve wellcontrolled BP. If BP is not well-Clinically significant increase in controlled within 2 weeks, DBP of 20 mmHg (but still below consider referral to a specialist 100 mmHg). and go to scenario (B).

| Management and Trametinib Dose Modification for Hypertension | | |
|---|---|---|
| Event | Management Guideline | Dose Modification |
| (Scenario B) Asymptomatic SBP ≥160 mmHg, or DBP ≥100 mmHg, or Failure to achieve well-controlled BP within 2 weeks in Scenario A. | <ul> <li>Adjust current or initiate new<br/>antihypertensive medication(s).</li> <li>Titrate antihypertensive<br/>medication(s) during the next 2<br/>weeks to achieve well-<br/>controlled BP.</li> </ul> | <ul> <li>Interrupt trametinib if clinically indicated.</li> <li>Once BP is well-controlled, restart trametinib reduced by one dose level.<sup>a</sup></li> </ul> |
| (Scenario C) Symptomatic hypertension or Persistent SBP ≥ 160 mmHg, or DBP ≥ 100 mmHg, despite antihypertensive medication and dose reduction of trametinib | <ul> <li>Adjust current or initiate new antihypertensive medication(s).</li> <li>Titrate antihypertensive medication(s) during the next 2 weeks to achieve well-controlled BP.</li> <li>Referral to a specialist for further evaluation and follow-up is recommended.</li> </ul> | Interrupt trametinib. Once BP is well-controlled, restart trametinib reduced by one dose level. <sup>a</sup> |
| (Scenario D) Refractory hypertension unresponsive to above interventions or hypertensive crisis. | Continue follow-up per protocol. | Permanently discontinue trametinib. |

a. Escalation of trametinib to previous dose level can be considered if BPs remain well controlled for 4 weeks after restarting of trametinib. Approval from the subprotocol Study Chair is required.

# 3.4.4 Guidelines for Visual Changes

Trametinib is known to be associated with visual adverse events. An ophthalmologist should be consulted if changes in vision develop. However, if the visual changes are clearly unrelated to study treatment (e.g., allergic conjunctivitis), then monitor closely as it may be reasonable to defer ophthalmic examination. Special attention should be given to retinal findings (e.g., retinal pigment epithelial detachment (RPED) or retinovascular abnormalities (i.e., branch or central retinal vein occlusions [RVO]).

The ophthalmology exam will include best corrected visual acuity, visual field examination, tonometry, slit lamp biomicroscopic examination, and indirect fundoscopy. Optical coherence tomography is recommended at scheduled visits and if retinal abnormalities are suspected. Other types of ancillary testing including visual field examination, fundus photography, and fluorescein angiography may also be indicated as determined by clinical exam.

Guidelines regarding event management and dose reduction for visual changes considered to be related to study treatment are provided in Tables 4 and 5.

Management and Dose Modification Guidelines for Visual Changes and/or Table 4 **Ophthalmic Examination Findings** 

**EAY131-S2** 

| CTCAE<br>Grade <sup>a,c</sup> | Adverse Event<br>Management | Action and Dose Modification |
|---|---|---|
| Grade 1 <sup>b</sup> | Consult<br>ophthalmologist<br>within 7 days of<br>onset | <ul> <li>If dilated fundus examination cannot be performed within 7 days of onset, interrupt trametinib until RPED and RVO can be excluded by retina specialist/ophthalmologist.</li> <li>If RPED and RVO excluded, continue/or restart trametinib at same dose level</li> <li>If RPED suspected or diagnosed: see RPED dose modification table below (following this table); report as SAE.</li> <li>If RVO diagnosed: Permanently discontinue trametinib and report as SAE.</li> </ul> |
| Grade 2 and<br>Grade 3 | Consult<br>ophthalmologist<br>immediately | <ul> <li>Hold trametinib</li> <li>If RPED and RVO excluded, restart trametinib at same dose level after visual AE is ≤ grade 1. If no recovery within 4 weeks, discontinue trametinib.</li> <li>If RPED diagnosed, see RPED dose modification table below; report as SAE.</li> <li>If RVO diagnosed: Permanently discontinue trametinib and report as SAE.</li> </ul> |
| Grade 4 | <ul> <li>Consult ophthalmologist immediately</li> <li>Report as SAE</li> </ul> | <ul> <li>Hold trametinib</li> <li>If RPED and RVO excluded, may restart trametinib at same or reduced dose after discussion with the subprotocol Study Chair</li> <li>If RVO or RPED diagnosed, permanently discontinue trametinib</li> </ul> |

Abbreviations: RPED = retinal pigment epithelial detachment; CTCAE = Common Terminology Criteria for Adverse Events;

RVO= retinal vein occlusion; SAE = serious adverse event

- a. Refers to CTCAE Version 4.0 'Eye disorders Other, specify'
- b. If visual changes are clearly unrelated to study treatment (e.g., allergic conjunctivitis), monitor closely but ophthalmic examination is not required.
- c. Refers to CTCAE Version 4.0 'Retinopathy'

Recommended dose modifications for trametinib for retinal pigment epithelial Table 5 detachments (RPED)a

| CTCAE Grade | Action and Dose Modification |
|---|---|
| Grade 1 RPED (Asymptomatic; clinical or diagnostic observations only) | Continue treatment with retinal evaluation monthly until<br>resolution. If RPED worsens follow instructions below |
| Grade 2-3 RPED (Symptomatic with mild to moderate decrease in visual acuity; limiting instrumental ADL) | <ul> <li>Interrupt trametinib</li> <li>Retinal evaluation monthly</li> <li>If improved to ≤ Grade 1, restart trametinib at lower dose (reduced by 0.5 mg) or discontinue in patients taking trametinib 1 mg daily</li> </ul> |
| | <ul> <li>If no recovery within 4 weeks, permanently discontinue trametinib</li> </ul> |

# 3.4.5 Pneumonitis Management Guidelines

Pneumonitis has been observed in subjects receiving trametinib. To reduce the risk of pneumonitis, subjects will be monitored closely for symptoms, evaluated with imaging and functional tests. Dose modification and supportive care guidelines for pneumonitis are described (see Table 6).

Table 6 Pneumonitis Guidelines for Trametinib

| CTCAE<br>Grade | Adverse Event Management | Action and Dose Modification |
|---|---|---|
| Grade 1 | <ul> <li>CT scan (high-resolution with lung windows) recommended</li> <li>Clinical evaluation and laboratory work-up for infection</li> <li>Monitoring of oxygenation via pulse-oximetry recommended</li> <li>Consultation with pulmonologist recommended</li> </ul> | Continue trametinib at current dose |
| Grade 2 | <ul> <li>CT scan (high-resolution with lung windows) recommended</li> <li>Clinical evaluation and laboratory work-up for infection</li> <li>Consult pulmonologist</li> <li>Pulmonary function tests -if &lt; normal, repeat every 8 weeks until ≥ normal</li> <li>Bronchoscopy with biopsy and/or BAL recommended</li> <li>Symptomatic therapy including corticosteroids if clinically indicated</li> </ul> | <ul> <li>Interrupt trametinib until recovery to grade ≤ 1</li> <li>Restart treatment with trametinib reduced by one dose level</li> <li>Escalation to previous dose level after 4 weeks and consultation with the subprotocol Study Chair possible</li> <li>If no recovery to grade ≤ 1 within 2 weeks, permanently discontinue trametinib</li> </ul> |
| Grade 3 | Same as Grade 2 | <ul> <li>Interrupt trametinib until recovery to grade ≤1</li> <li>After consultation with the subprotocol Study Chair, treatment with trametinib may be restarted reduced by one dose level</li> <li>If no recovery to grade ≤ 1 within 2 weeks, permanently discontinue trametinib</li> </ul> |
| Grade 4 | Same as Grade 2 | Permanently discontinue trametinib |

Abbreviations: BAL= bronchioalveolar lavage; CT = computed tomography; CTCAE = Common Terminology Criteria for Adverse Events

EAY131-S2 Version Date: August 19, 2020

Dose Modifications for Trametinib and supportive care 3.5

Rev. 12/16

#### **Trametinib Dose Modification for Liver Chemistry Changes** 3.5.1

#### Trametinib Dose Modification for Liver Function Test Abnormalities Table 7:

| Event Treatment modifications and assessment/monitoring | |
|---|---|
| ALT ≥ 3x ULN but < 5x ULN and TB < 2x ULN, without symptoms considered related to liver injury or hypersensitivity and who can be monitored weekly for 4 weeks | <ul> <li>May continue study drug.</li> <li>Report as SAE if CTEP-AERS reporting criteria is met.</li> <li>If liver chemistry stopping criteria are met any time, proceed as described below.</li> <li>MONITORING:</li> <li>Repeat LFT (ALT, AST, ALK, bilirubin) until they return to normal/baseline or stabilise (LFT may be every 2 weeks after 4 weeks if ALT &lt; 3x ULN and TB &lt; 2 ULN). If baseline ALT and Tbili already meet these criteria, then monitoring is required only if ALT or TB rises after initiation of study therapy.</li> </ul> |
| Criteria for discontinuing study drug: When any of the liver stopping criteria below is met, discontinue trametinib 1. ALT≥3xULN and bilirubin ≥ 2x ULN or >35% direct bilirubin ¹.² 2. ALT≥ 3xULN and INR >1.5, if INR measured² (INR threshold does not apply if subject is on anticoagulant) 3. ALT≥ 5x ULN 4. ALT≥ 3x ULN persists for ≥ 4 weeks. However, if ALT was elevated 3-5x at baseline due to liver mets, then this criteria should not be used for treatment discontinuation UNLESS the ALT improves to < 3x ULN and then subsequently rises. 5. ALT≥ 3x ULN and cannot be monitored weekly for 4 weeks. However, if ALT was elevated 3-5x at baseline due to liver mets, then this criteria should not be used for treatment discontinuation UNLESS the ALT improves to < 3x ULN and then subsequently rises. 6. ALT≥ 3x ULN associated with symptoms³ (new or worsening) believed to be related to liver injury or | <ul> <li>Immediately discontinue study treatment.</li> <li>Do not restart/rechallenge unless approved by the subprotocol Study Chair. [</li> <li>Report as SAE if: 1) CTEP-AERS reporting criteria are met, or 2) patients meet criteria 1-2.</li> <li>Perform liver event ASSESSMENT AND WORKUP (see below).</li> <li>Monitor the subject until liver chemistries resolve, stabilize, or return to baseline (see MONITORING below).</li> <li>If applicable, provide details on required follow up assessments (e.g., follow up for overall survival or disease recurrence or progression). [Do not include for single-dose studies]</li> <li>MONITORING:</li> <li>In patients stopping for criteria 1-2 (with abnormal TB and INR, indicating potentially more significant liver toxicities):</li> <li>Repeat liver chemistries (ALT, AST, ALK, bilirubin) and perform liver event follow-up assessments within 24 hours.</li> <li>Monitor subjects twice weekly until LFT return to normal/baseline or stabilize.</li> <li>A specialist or hepatology consultation is recommended. In patients stopping for criteria 2-6:</li> <li>Repeat LFT and perform liver event follow up assessments within 24-72 hrs</li> <li>Monitor subjects weekly until LFTs return to normal/baseline or stabilize.</li> <li>ASSESSMENT and WORKUP:</li> <li>Viral hepatitis serology.<sup>4</sup></li> <li>Serum CPK and LDH.</li> <li>Fractionate bilirubin, if total bilirubin ≥ 2x ULN.</li> <li>CBC with differential to assess eosinophilia.</li> <li>Record clinical symptoms of liver injury, or hypersensitivity on AE</li> </ul> |
| hypersensitivity | CRF. • Record concomitant medications (including acetaminophen, herbal |

| Event | Treatment modifications and assessment/monitoring |
|---|---|
| | remedies, other over the counter medications). |
| | Record alcohol use. |
| | Additional work up for patient stopping for criteria 1-2 (with abnormal TB and INR, indicating potentially more significant liver toxicities): |
| | <ul> <li>Anti-nuclear antibody, anti-smooth muscle antibody, Type 1 anti-<br/>liver kidney microsomal antibodies, and quantitative total<br/>immunoglobulin G (lgG or gamma globulins).</li> </ul> |
| | Serum acetaminophen adduct HPLC assay (in subjects with likely acetaminophen use in the preceding). |
| | <ul> <li>If there is underlying chronic hepatitis B (e.g. positive hepatitis B<br/>surface antigen): quantitative hepatitis B DNA and hepatitis delta<br/>antibody.<sup>5</sup></li> </ul> |
| | Liver imaging (ultrasound, MRI, CT) and /or liver biopsy. |

# Footnotes:

- 1. Serum bilirubin fractionation should be performed if testing is available. If serum bilirubin fractionation testing is unavailable, record presence of detectable urinary bilirubin on dipstick, which indicates direct bilirubin elevations and suggesting liver injury.
- 2. All events of ALT≥3xULN and bilirubin ≥2xULN (>35% direct bilirubin) or ALT ≥3x ULN and INR > 1.5 (if INR measured) may indicate severe liver injury (possible "Hy's Law"). INR measurement is not required, and the threshold value stated will not apply to subjects receiving anticoagulants.
- 3. New or worsening symptoms believed to be related to liver injury (such as fatigue, nausea, vomiting, right upper quadrant pain or tenderness, or jaundice) or believed to be related to hypersensitivity (such as fever, rash or eosinophilia)
- 4. Includes: Hepatitis A IgM antibody; Hepatitis B surface antigen and Hepatitis B Core Antibody (IgM); Hepatitis C RNA; Cytomegalovirus IgM antibody; Epstein-Barr viral capsid antigen IgM antibody (or if unavailable, obtain heterophile antibody or monospot testing); Hepatitis E IgM antibody
- 5. If hepatitis delta antibody assay cannot be performed, it can be replaced with a PCR of hepatitis D RNA virus (where needed) (Le Gal *et al.*, 2005).

# 3.5.2 Guidelines for Prolonged QTc

Guidelines for dose modification and stopping criteria due to QT c-prolongation are provided (see Table 8).

# Table 8 Withholding and Stopping Criteria for QTc-Prolongation

| QTc-Prolongation <sup>a</sup> | Action and Dose Modification |
|---|---|
| • QTcB ≥ 501 msec, or | Interrupt all study treatments until QTcB prolongation resolves to grade 1 or baseline |
| <ul><li>Uncorrected QT &gt; 600 msec, or</li></ul> | <ul> <li>Test serum potassium, calcium, phosphorus and magnesium. If<br/>abnormal correct per routine clinical practice to within normal limits.</li> </ul> |
| • QTcB > 530 msec | Review concomitant medication usage for a prolonged QTc. |
| for subjects with bundle branch block | Restart at current dose level <sup>b</sup> |
| | <ul> <li>If event does not resolve or recurs after restarting, permanently<br/>discontinue study treatments.</li> </ul> |

Abbreviations: msec = milliseconds; QTcB = QT interval on electrocardiogram corrected using the Bazett's formula

- A: Based on average QTc value of triplicate ECGs. For example, if an ECG demonstrates a prolonged QT interval, obtain two or more ECGs over a brief period, and then use the averaged QTc values of the three ECGs to determine if study treatments should be interrupted or discontinued.
- B: If the QTc prolongation resolves to grade 1 or baseline, the subject may resume study treatment if the investigator and the subprotocol Study Chair agree that the subject will benefit from further treatment.

Rev. 12/16

# 3.5.3 **Guidelines for Rash**

Rash is a frequent AE observed in subjects receiving trametinib (see the Investigator's Brochures [4]] for more information). Recommendations for supportive care and guidelines for dose modifications for rash are based on experience with other MEK inhibitors and EGFR inhibitors [26, 27] and are provided (see Table 9 and Table 10.

The institutional standards for the management of skin-related AEs can differ from these guidelines. In this case, best clinical judgment should be applied and a consultation with the subprotocol Study Chair may be required.

Table 9 Guidelines for Supportive Care of Rash

| Type of Care | Action |
|---|---|
| Prevention/Prophylaxis <sup>a</sup> | <ul> <li>Avoid unnecessary exposure to sunlight</li> <li>Apply broad-spectrum sunscreen (containing titanium dioxide or zinc oxide) with a skin protection factor (SPF)≥15 at least twice daily.</li> <li>Use thick, alcohol-free emollient cream (e.g., glycerine and cetomacrogol cream) on dry areas of the body at least twice daily.</li> <li>Topical steroids and/or antibiotics should be applied at least twice daily starting on Day 1 of study treatment, to body areas such as face, chest, and upper back.</li> <li>Use mild-strength topical steroid (hydrocortisone 1% cream) and/or</li> </ul> |
| | topical antibiotic (e.g., clindamycin) or oral antibiotics (e.g., doxycycline 100 mg BID, minocycline 100 mg BID) |
| Symptomatic Care <sup>b</sup> | <ul> <li>Pruritic lesions: cool compresses and oral antihistamine therapies</li> <li>Fissuring lesions: Monsel's solution, silver nitrate, or zinc oxide cream</li> <li>Desquamation: thick emollients and mild soap</li> </ul> |
| | <ul> <li>Paronychia: antiseptic bath, local potent corticosteroids in addition<br/>to oral antibiotics; if no improvement, consult dermatologist or<br/>surgeon</li> </ul> |
| | <ul> <li>Infected lesions: appropriate bacterial/fungal culture-driven<br/>systemic or topical antibiotics</li> </ul> |

Abbreviations: BID = twice daily; SPF = sun protection factor

- a. Rash prophylaxis is recommended for the first 6 weeks of study treatment
- b. Subjects who develop rash/skin toxicities should be seen by a qualified physician and should receive evaluation for symptomatic/supportive care management

Guidelines for management and dose reduction for rash considered to be related to study treatment are provided (see Table 10).

Table 10 Management and Dose Modification Guidelines for Rash

| CTCAE<br>Grade | Adverse Event Management | Action and Dose Modification |
|---|---|---|
| Grade 1 | <ul> <li>Initiate prophylactic and<br/>symptomatic treatment<br/>measures<sup>a</sup></li> <li>Use moderate strength topical<br/>steroid<sup>b</sup></li> <li>Reassess after 2 weeks</li> </ul> | Continue study treatment If rash does not recover to baseline within 2 weeks despite best supportive care, reduce trametinib by one dose level <sup>c</sup> |
| Grade 2 | <ul> <li>Initiate prophylactic and<br/>symptomatic treatment<br/>measures</li> <li>Use moderate strength topical<br/>steroid<sup>b</sup></li> <li>Reassess after 2 weeks</li> </ul> | <ul> <li>Reduce trametinib by one dose level</li> <li>If rash recovers to ≤ grade 1 within 2 weeks, increase dose to previous dose level</li> <li>If no recovery to ≤ grade 1 within 2 weeks, interrupt study treatment until recovery to ≤ grade 1</li> <li>Restart trametinib at reduced dose level<sup>c</sup></li> </ul> |
| Grade≥3 | <ul> <li>Use moderate strength topical steroids<sup>b</sup> PLUS oral methylprednisolone dose pack</li> <li>Consult dermatologist</li> </ul> | <ul> <li>Interrupt trametinib until rash recovers to grade ≤ 1</li> <li>Restart<sup>c</sup> trametinib reduced by one dose level<sup>d</sup></li> <li>If no recovery to grade ≤ 2 within 2 weeks, permanently discontinue trametinib</li> </ul> |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events

- a. Rash prophylaxis is recommended for the first 6 weeks of study treatment
- b. Moderate-strength topical steroids: hydrocortisone 2.5% cream or fluticasone prioprionate 0.5% cream
- c. Approval of subprotocol Study Chair is required to restart study treatment after > 2 weeks of interruption.
- d. Escalation of study treatment to previous dose level may be considered if no rash is evident 4 weeks after restarting study treatment

Rev. 12/16

# 3.5.4 Guidelines for Diarrhea

Episodes of diarrhea have occurred in subjects receiving trametinib (see the Investigator Brochures [4] for more information). Other, frequent causes for diarrhea including concomitant medications (e.g., stool softeners, laxatives, antacids, etc.), infections by *C. difficile* or other pathogens, partial bowel obstruction, etc., should be clinically excluded.

Guidelines regarding management and dose reduction for diarrhea considered to be related to trametinib by the investigator are provided (see Table 11).
Table 11 Management and Dose Modification Guidelines for Diarrhea

EAY131-S2

| CTCAE Grade | Adverse Event Management | Action and Dose Modification |
|---|---|---|
| Uncomplicated<br>Diarrhea <sup>a</sup><br>Grade 1 or 2 | <ul> <li><u>Diet:</u> stop all lactose containing products; eat small meals, BRAT-diet (banana, rice, apples, toast) recommended</li> <li><u>Hydration:</u> 8-10 large glasses of clear liquids per day (e.g., Gatorade or broth)</li> <li><u>Loperamide<sup>c</sup>:</u> initially 4 mg, followed by 2 mg every four hours or after every unformed stool; maximum 16 mg/day. Continue until diarrhea free for 12 hours</li> <li><u>Diarrhea &gt; 24</u>h: loperamide 2 mg every two hours; maximum 16 mg/day. Consider adding oral antibiotics</li> <li><u>Diarrhea &gt; 48h:</u> loperamide 2 mg every two hours; maximum 16 mg/day. Add budesonide</li> </ul> | <ul> <li>Continue trametinib</li> <li>If diarrhea is grade 2 for &gt; 48h, interrupt trametinib until diarrhea resolves to grade ≤1</li> <li>Restart trametinib at the same dose level</li> <li>If treatment delay is &gt; 14 days, discontinue trametinib.</li> </ul> |
| | or other second-line therapies (otreotide, or tincture of opium) and oral antibiotics | |
| Uncomplicated<br>Diarrhea <sup>a</sup><br>Grade 3 or 4<br>Any<br>Complicated<br>Diarrhea <sup>b</sup> | <ul> <li>Clinical evaluation mandatory</li> <li>Loperamide<sup>c</sup>: initially 4 mg, followed by 2 mg every four hours or after every unformed stool; maximum 16 mg/day. Continue until diarrhea free for 12 hours</li> <li>Oral antibiotics and second-line therapies if clinically indicated</li> <li>Hydration: intravenous fluids if clinically indicated</li> <li>Antibiotics (oral or intravenous) if clinically indicated</li> </ul> | <ul> <li>Interrupt trametinib until diarrhea resolves to grade ≤1</li> <li>Restart with trametinib reduced by one dose level<sup>d</sup></li> <li>If 3 dose reductions of study treatment are clinically indicated, permanently discontinue trametinib</li> </ul> |
| | <ul> <li>Intervention should be continued until the subject is diarrhea free for ≥ 24 hours</li> <li>Intervention may require hospitalization for subjects at risk of life-threatening complications</li> </ul> | |

Abbreviation: CTCAE = Common Terminology Criteria for Adverse Events

- **Uncomplicated diarrhea** defined by the absence of symptoms such as, cramping, nausea/vomiting ≥ grade 2, decreased performance status, pyrexia, sepsis, neutropenia grade ≥ 3, frank bleeding, and/or dehydration requiring intravenous fluid substitution
- Complicated diarrhea defined by the presence of symptoms such as, cramping, nausea/vomiting ≥ grade 2, decreased performance status, pyrexia, sepsis, neutropenia grade ≥ 3, frank bleeding, and/or dehydration requiring intravenous fluid substitution
- c. Loperamide should be made available prior to start of study treatment so loperamide administration can begin at the first signs of diarrhea
- Escalation of trametinib to previous dose level is allowed after consultation with the Subprotocol Study Chair and in the absence of another episode of complicated or severe diarrhea in the 4 weeks subsequent to dose reduction.

Rev. 12/16

3.5.5 Trametinib Dose Modification for Toxicities Not Specified in **Subsequent Sections** 

## Table 12 Trametinib Treatment Modification for Clinically Significant Toxicities Deemed Related to Trametinib

(This section is <u>not</u> for specific AEs such as hypertension, rash, ejection fraction changes, pneumonitis, diarrhea, liver chemistry, or visual changes. Refer to <u>other</u> sections for these specific AEs).

| CTCAE v4 Grade | Management Guideline | Dose Modification |
|---|---|---|
| Grade 1 | Monitor as clinically | Continue trametinib at current dose level. |
| Grade 2 (tolerable) | indicated. Provide supportive care according to institutional standards. | baseline. |
| | | Upon resolution, restart treatment at current dose level. |
| Grade 2 (intolerable) and | | Interrupt treatment until resolution to grade 1 or baseline. |
| Grade 3 | | Upon resolution to baseline or grade 1, restart with one level of dose reduction. |
| | | <ul> <li>If the Grade 3 toxicity recurs, interrupt trametinib;</li> <li>When toxicity resolves to Grade 1 or baseline, restart<br/>trametinib reduced by another dose level.</li> </ul> |
| Grade 4 | | If event resolves to grade 1 or baseline discuss potential continuation of trametinib with the subprotocol Study Chair; if continuation of treatment agreed then restart trametinib at dose <b>reduced by one dose level</b> . |
| | | If event does not resolve, permanently discontinue trametinib. |

Trametinib should be discontinued if treatment delay is ≥14 days due to toxicities. If the investigator concludes that continued trametinib will benefit a patient, the subprotocol Study Chair may be consulted for the possibility of resuming trametinib, provided that toxicities have resolved to baseline or grade 1.

### 3.6 Supportive Care

All supportive measures consistent with optimal patient care will be given throughout the study.

### 3.7 Duration of Agent-specific treatment

In the absence of treatment delays due to adverse event(s), treatment may continue until one of the following criteria applies:

- Extraordinary Medical Circumstances: If at any time the constraints of this
  protocol are detrimental to the patient's health, protocol treatment should be
  discontinued. In this event submit forms according to the instructions in the
  MATCH Forms Packet.
- Patient withdraws consent.
- Patient experiences unacceptable toxicity.
- Non-protocol therapies are administered.
- Disease Progession

### 3.8 Duration of Follow-Up

Refer to the MATCH Master Protocol for specifics on the duration of follow-up.

### **Study Parameters** Rev. 12/16 **4.**

#### 4.1 Therapeutic Parameters for Trametinib Treatment

In addition to the study parameters listed in the main screening protocol, the below parameters must also be NOTE:

performed for patients receiving Trametinib treatment.

NOTE: All assessments required prior to registration to treatment should be done ≤ 4 weeks prior to registration to

Steps 1, 3, 5, 7, excluding the radiologic evaluation and electrocardiogram (ECG).

| | Prior to | Treatment | | End of | Fallow |
|---|---|---|---|---|---|
| Test/Assessment | Registration to<br>Treatment | Every Cycle, prior to treatment | Every 2<br>Cycles | End of Treatment | Follow<br>Up <sup>F</sup> |
| H&P, Weight, Vital signs <sup>A</sup> | Х | X <sub>1</sub> | | | Х |
| Performance status | Х | X <sub>1</sub> | | | Х |
| CBC w/diff, plts <sup>B</sup> | Х | X <sub>1</sub> | | | Х |
| Serum chemistry <sup>B</sup> | Х | X <sub>1</sub> | | | Х |
| Radiologic evaluation <sup>D</sup> | Х | | XD | | X <sup>F</sup> |
| β-HCG <sup>c</sup> | Х | | | | |
| Toxicity Assessment <sup>G</sup> | Х | X | | Х | X <sup>F</sup> |
| Pill Count/Diary <sup>H</sup> | | X | | Х | |
| ECG <sup>K</sup> | Х | Χ <sup>L</sup> | | | |
| Echo cardiogram or Nuclear Study <sup>L</sup> | Х | Χ <sup>L</sup> | | | |
| Eye exam | Х | Χı | | | |
| Tumor biopsy and blood sample for MATCH Master Protocol <sup>E</sup> | | | Χ | Х | |

Rev. 3/17

- A. History and physical, including vital signs and weight at the start of each cycle (up to 3 days before start of new cycle).
- B. Albumin, alkaline phosphatase, total bilirubin, bicarbonate, BUN, calcium, creatinine, glucose, phosphorus, potassium, SGOT[AST], SGPT[ALT], sodium, magnesium, and serum tumor markers (including LDH, PSA if appropriate). For eligibility purposes, participants with creatinine levels above institutional normal, Cockcroft-Gault will be used to calculate creatinine clearance. CBC w/diff, platelets and serum chemistries should be performed on cycle 1, day 1 (or up to 7 days prior), and at the start of each subsequent cycle (up to 3 days before start of new cycle). CBC with differential will be performed more frequently in patients with grade 4 neutropenia or thrombo cytopenia until resolution to ≤ grade 3. CBC and serum chemistries are only required in follow-up until values return to pre-treatment levels or until progressive disease.
- C. Blood pregnancy test (women of childbearing potential) required prior to beginning treatment.

D. Disease measurements are repeated every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until PD or start of another MATCH treatment step. The baseline evaluation should be performed as closely as possible to the beginning of treatment and never more than 6 weeks before registration to treatment step. For multiple myeloma patients, please refer to Section 6.4 of the MATCH Master Protocol for additional information on myeloma response criteria and the required disease assessments. Documentation (radiologic) must be provided for patients removed from study for progressive disease.

Rev. 3/17 Rev. Add13

- E. Additional blood specimens and/or biopsies are to be submitted from consenting platients per Section 9.3.2 of the MATCH Master Protocol. Submit at the following time points, as applicable:
  - Blood specimens are to be submitted at the end of Cycle 2 (prior to start of Cycle 3 treatment). If patient progresses or treatment is discontinued prior to Cycle 3, collect the blood at that time instead. On-treatment kits for blood sample collections will be automatically shipped to sites upon registration to the treatment step.
  - Screening biopsies for additional aMOI assessments after registration to appropriate screening step, if applicable (Step 2 or Step 4).
  - At end of all MATCH study treatments, blood specimens and/or research biopsy after consent and registration to Step 8 Please refer to Section 4 of the MATCH Master Protocol to determine whether the patient proceeds to the next screening step or to follow-up (with a potential end of treatment biopsy for research purposes on Step 8). Samples are to be submitted as outlined in Section 9 of the MATCH

Master Protocol. To order Step 2/4 Screening or Step 8 kits, complete the EAY131 Collection and Shipping Kit Order Form (See Appendix XII of the MATCH Master Protocol) and fax to 713-563-6506.

- F. Every 3 months if patient is < 2 years from study entry, and every 6 months for year 3. Toxicity assessments and radiologic evaluations are not required to be done during Follow Up if progression has been previously reported; however if an adverse event occurs post treatment that meets the SAE reporting requirements, it still must be reported via CTEP-AERS, even if progression has occurred.
- G. Site personnel should evaluate for toxicity and discuss treatment compliance with the patient in order to ensure the medication is taken correctly; this evaluation may be conducted by telephone or in person. The Toxicity Assessment is not required prior to Cycle 1, but is required every subsequent cycle.
- H. The pill calendar will be collected at the end of every cycle. The Pill Count/Diary is not required prior to Cycle 1, but is required every subsequent cycle.
- As clinically indicated.
- J. For Cycle 1, if the following tests/assessments occurred within 7 days of Day 1, they do not need to be repeated at this time point: H&P, Weight, Vital signs; Performance Status; CBC w/diff, plts; Serum chemistry; Concomitant Medications.
- K. Within 8 weeks of treatment assignment.
- L. Cardiac monitoring with ECG and either ECHO or Nuclear Study (MUGA or First Pass) is needed at week 5, week 13, and every 12 weeks thereafter unless clinically indicated sooner. The same modality should be used at baseline and thereafter.

### Rev. Add13 5. Rev. Add25

## **Drug Formulation and Procurement**

This information has been prepared by the ECOG-ACRIN Pharmacy and Nursing Committees.

## **Availability**

NO STARTER SUPPLIES MAY BE ORDERED. Subjects must be enrolled and assigned to the treatment subprotocol prior to submitting the clinical drug request to PMB.

Drug Ordering: NCI supplied agents may be requested by eligible participating Investigators (or their authorized designee) at each participating institution. Pharmaceutical Management Branch (PMB) policy requires that drug be shipped directly to the institution where the patient is to be treated. PMB does not permit the transfer of agents between institutions (unless prior approval from PMB is obtained – see general information) The CTEP-assigned protocol number must be used for ordering all CTEPsupplied investigational agents. The eligible participating investigators at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA Form 1572 (Statement of Investigator), NCI Biosketch, Agent Shipment Form, and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP-supplied investigational agents for the study should be ordered under the name of one lead investigator at that institution.

Submit agent requests through the PMB Online Agent Order Processing (OAOP) application (https://ctepcore.nci.nih.gov/OAOP). Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account (https://ctepcore.nci.nih.gov/iam/) and the maintenance of an "active" account status, a "current" password, and an active person registration status.

## NCI Supplied Agent(s) - General Information

Questions about drug orders, transfers, returns, or accountability should be addressed to the PMB by calling 240-276-6575 Monday through Friday between 8:30 AM and 4:30 PM Eastern Time or email <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> anytime.

Drug Returns: All undispensed drug supplies should be returned to the PMB. When it is necessary to return study drug (e.g., sealed bottles remaining when PMB sends a stock recovery letter), investigators should return the study drug to the PMB using the NCI Return Agent Form available on the NCI home page (http://ctep.cancer.gov).

Drug Accountability: The investigator, or a responsible party designated by the investigator, must maintain a careful record of the receipt, disposition, and return of agent received from the PMB using the NCI Investigational Agent Accountability Record Form for Oral Agents available on the NCI home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>). Maintain separate NCI Investigational Agent Accountability Records for each agent, strength. formulation and ordering investigator.

Investigator Brochure Availability: The current versions of the IBs for PMB-supplied agents will be accessible to site investigators and research staff through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account and the maintenance of an "active" account status, a "current" password, and active person registration status. Questions about IB access may be directed to the PMB IB coordinator at <a href="mailto:IBCoordinator@mail.nih.gov">IBCoordinator@mail.nih.gov</a>.

Rev. 12/16

Rev. 3/17

### 5.1 Trametinib dimethyl sulfoxide (NSC 763093)

#### 5.1.1 Other Names

Trametinib, GSK1120212B, TMT212-NXA, JTP-74057, JTP-78296, JTP-75303, Mekinist®

#### 5.1.2 Classification

MFK inhibitor

Rev. 12/16

#### 5.1.3 Mode of Action

Trametinib dimethyl sulfoxide is a reversible, highly selective, allosteric inhibitor of mitogen-activated extracellular signal regulated kinase 1 (MEK1) and MEK2. Tumor cells commonly have hyperactivated extracellular signal-related kinase (ERK) pathways in which MEK is a critical component. Trametinib dimethyl sulfoxide inhibits activation of MEK by RAF kinases and MEK kinases.

#### 5.1.4 Storage and Stability

**Storage:** Store tablets at 2°C -8°C (36° F to 46° F) in the original bottle and dispense unopened bottles. Do not open bottles or repackage tablets or remove desiccant. Bottles should be protected from light and moisture.

If a storage temperature excursion is identified, promptly return trametinib to 2°C -8°C and guarantine the supplies. Provide a detailed report of the excursion (including documentation of temperature monitoring and duration of the excursion) to PMBAfterHours@mail.nih.gov for determination of suitability.

**Stability:** Stability studies are ongoing. Tablets are only stable for 32 days once bottle has been opened. If multiple bottles are dispensed to a patient in the same visit, please advise the patient to open only one bottle at a time.

**Storage:** Refer to the package label for expiration.

### 5.1.5 **Dose Specifics**

Trametinib will be given continuous dosing 2mg daily.

5.1.6 Preparation

> Novartis supplies and CTEP, NCI, DCTD distributes trametinib as 0.5 mg and 2 mg (as free base) tablets. Each investigationally-labeled bottle contains 32 tablets with a desiccant.

The tablet core contains mannitol, microcrystalline cellulose. hypromellose, croscarmellose sodium, magnesium stearate (nonanimal), colloidal silicon dioxide and sodium lauryl sulfate.

- 0.5 mg tablets are yellow, modified oval, biconvex and film-coated. Agueous film coating consists of hypromellose, titanium dioxide, polyethylene glycol, iron oxide yellow.
- 2 mg tablets are pink, round, biconvex and film-coated. Aqueous film coating consists of hypromellose, titanium dioxide, polyethylene glycol, polysorbate 80, iron oxide red.

Rev. 12/16

Rev.5/16

5.1.9 Side Effects

See Section 3.3 for side effects.

5.1.10 Nursing/Patient Implications

Advise women study participants of reproductive potential to use effective contraception while receiving study treatment and for 4 months after the last dose of trametinib. Advise women not to breastfeed while receiving study treatment and for 4 months after the last dose of trametinib. Advise men study participants to use barrier contraception and not to father a child while taking study treatment and for 4 months after the last dose of trametinib.

### 6. Translational Studies

Please refer to the MATCH Master Protocol for information on the Translational Studies.

### 7. References

Ambrosini, G., Musi, E., Ho, A. L., De Stanchina, E., and Schwartz, G. K. (2013). Inhibition of mutant GNAQ signaling in uveal melanoma induces AMPK-dependent autophagic cell death. Molecular cancer therapeutics 12, 768-76.

Ambrosini, G., Pratilas, C. A., Qin, L. X., Tadi, M., Surriga, O., Carvajal, R. D., and Schwartz, G. K. (2012). Identification of unique MEK-dependent genes in GNAQ mutant uveal melanoma involved in cell growth, tumor cell invasion, and MEK-resistance. Clin Cancer Res 18 1-10.

Ars E, Kruyer H, Morell M, et al. Recurrent mutations in the NF1 gene are common among neurofibromatosis type 1 patients. J Med Genet 2003;40:e82.

Balagula, Y., K. Barth Huston, K.J. Busam, *et al.* (2010). Dermatologic side effects associated with the MEK 1/2 inhibitor selumetinib (AZD6244, ARRY-142886). *Invest New Drugs.* 29:1114-1121.

Bekaii-Saab, T., M.A. Phelps, X. Li, *et al.* (2011). Multi-institutional phase II study of selumetinib in patients with metastatic biliary cancers. *J Clin Oncol.* 29:2357-2363.

Bendell, J., P. LoRusso, E. Kwak, *et al.* (2011). Clinical combination of the MEK inhibitor GDC-0973 and the PI3K inhibitor GDC-0941: A first-in-human phase Ib study in patients with advanced solid tumors. *AACR Meeting Abstracts*. Abstract LB-89.

Blumenschein, G.R., E.F. Smit, D. Planchard, *et al.* (2013). MEK114653: A randomized, multicenter, phase II study to assess efficacy and safety of trametinib (T) compared with docetaxel (D) in KRAS-mutant advanced non-small cell lung cancer (NSCLC). *J Clin Oncol.* 31:Abstract 8029.

Borthakur, G., J.M. Foran, T. Kadia, *et al.* (2010). GSK1120212, a MEK1/MEK2 inhibitor, demonstrates acceptable tolerability and preliminary activity in a dose rising trial In subjects with AML and other hematologic malignancies. *Blood (ASH Annual Meeting Abstracts)*. 116:Abstract 3281.

Brems H, Beert E, de Ravel T, Legius E. Mechanisms in the pathogenesis of malignant tumours in neurofibromatosis type 1. Lancet Oncol 2009;10:508-15.

Cancer Genome Atlas Research Network. Comprehensive genomic characterization defines human glioblastoma genes and core pathways. Nature. 2008;455:1061-8.

Carvajal, R. D., Sosman, J. A., Quevedo, F., Milhem, M. M., Joshua, A. M., Kudchadkar, R. R., Linette, G. P., Gajewski, T., Lutzky, J., Lawson, D. H., et al. (2013). Phase II study of selumetinib (sel) versus temozolomide (TMZ) in gnaq/Gna11 (Gq/11) mutant (mut) uveal melanoma (UM). J Clin Oncol 31, 2013 (suppl; abstr CRA9003).

Chang T, Krisman K, Theobald EH, et al. Sustained MEK inhibition abrogates myeloproliferative disease in Nf1 mutant mice. J Clin Invest 2013;123:335-9.

Cooper D, Upadhyaya M. The Germline Mutational Spectrum in Neurofibromatosis Type 1 and Genotype—Phenotype Correlations. In: Upadhyaya M, Cooper DN, eds. Neurofibromatosis Type 1: Springer Berlin Heidelberg; 2012:115-34.

Denayer E, de Ravel T, Legius E. Clinical and molecular aspects of RAS related disorders. J Med Genet 2008;45:695-703.

De Raedt T, Brems H, Wolkenstein P, et al. Elevated risk for MPNST in NF1 microdeletion patients. Am J Hum Genet 2003;72:1288-92.

Dilworth JT, Kraniak JM, Wojtkowiak JW, et al. Molecular targets for emerging anti-tumor therapies for neurofibromatosis type 1. Biochem Pharmacol 2006;72:1485-92.

Ebi, H., R.B. Corcoran, A. Singh, *et al.* (2011). Receptor tyrosine kinases exert dominant control over PI3K signaling in human KRAS mutant colorectal cancers. *J Clin Invest.* 121:4311-4321.

Engelman, J.A., L. Chen, X. Tan, *et al.* (2008). Effective use of PI3K and MEK inhibitors to treat mutant Kras G12D and PIK3CA H1047R murine lung cancers. *Nat Med.* 14:1351-1356.

Flaherty, K.T., C. Robert, P. Hersey, *et al.* (2012). Improved survival with MEK inhibition in BRAF-mutated melanoma. N Engl J Med. 367:107-114.

Frampton GM, Fichtenholtz A, Otto GA, et al. Development and validation of a clinical cancer genomic profiling test based on massively parallel DNA sequencing. Nat Biotechnol 2013;31:1023-31.

Gilmartin, A.G., M.R. Bleam, A. Groy, *et al.* (2011). GSK1120212 (JTP-74057) is an inhibitor of MEK activity and activation with favorable pharmacokinetic properties for sustained in vivo pathway inhibition. *Clin Cancer Res.* 17:989-1000.

Gopal, Y.N., W. Deng, S.E. Woodman, *et al.* (2010). Basal and treatment-induced activation of AKT mediates resistance to cell death by AZD6244 (ARRY-142886) in Brafmutant human cutaneous melanoma cells. *Cancer Res.* 70:8736-8747.

Gottfried ON, Viskochil DH, Fults DW, Couldwell WT. Molecular, genetic, and cellular pathogenesis of neurofibromas and surgical implications. Neurosurgery 2006;58:1-16; discussion 1-.

Griner, E. M., and Kazanietz, M. G. (2007). Protein kinase C and other diacylglycerol effectors in cancer. Nat Rev Cancer 7, 281-94.

Gursel DB, Connell-Albert YS, Tuskan RG, Anastassiadis T, Walrath JC, Hawes JJ, et al. Control of proliferation in astrocytoma cells by the receptor tyrosine kinase/PI3K/AKT signaling axis and the use of PI-103 and TCN as potential anti-astrocytoma therapies. Neuro Oncol. 2011;13:610-21.

Gutzmer R, Herbst RA, Mommert S, et al. Allelic loss at the neurofibromatosis type 1 (NF1) gene locus is frequent in desmoplastic neurotropic melanoma. Human genetics 2000;107:357-61.

Hodis E, Watson IR, Kryukov GV, et al. A landscape of driver mutations in melanoma. Cell 2012;150:251-63.

Hoeflich, K.P., C. O'Brien C, Z. Boyd, *et al.* (2009). In vivo antitumor activity of MEK and phosphatidylinositol 3-kinase inhibitors in basal-like breast cancer models. *Clin Cancer Res.* 15:4649-4664.

Holt, S. V., Logie, A., Odedra, R., Heier, A., Heaton, S. P., Alferez, D., Davies, B. R., Wilkinson, R. W., and Smith, P. D. (2012). The MEK1/2 inhibitor, selumetinib (AZD6244; ARRY-142886), enhances anti-tumour efficacy when combined with conventional chemotherapeutic agents in human tumour xenograft models. Br J Cancer 106, 858-66.

Hubbard, K. B., and Hepler, J. R. (2006). Cell signalling diversity of the Gqalpha family of heterotrimeric G proteins. Cell Signal 18, 135-50.

Infante, J.R., B.G. Somer, J.O. Park, *et al.* (2013). A randomized, double-blind, placebo-controlled trial of trametinib, a MEK inhibitor, in combination with gemcitabine for patients with untreated metastatic adenocarcinoma of the pancreas. *J Clin Oncol.* 30:Abstract 291.

Infante J.R., Fecher L.A., Falchook G.S., Nallapareddy S., *et al.* Safety, pharmacokinetic,, pharmacodynamics, and efficacy data for the oral MEK inhibitor trametinib; a phase I dose-escalation trial. Lancet Oncol 2012; 13(8): 773-81

Investigator's Brochure. (2012a). GSK1120212. *GlaxoSmithKline*. Version 04. September 5, 2012.

Investigator's Brochure. (2013). GSK1120212 (trametinib). *GlaxoSmithKline*. Version 05. September 25, 2013.

Ismat FA, Xu J, Lu MM, Epstein JA. The neurofibromin GAP-related domain rescues endothelial but not neural crest development in Nf1 mice. J Clin Invest 2006;116:2378-84.

Ivey, K., Tyson, B., Ukidwe, P., Mcfadden, D. G., Levi, G., Olson, E. N., Srivastava, D., and Wilkie, T. M. (2003). Galphaq and Galpha11 proteins mediate endothelin-1 signaling in neural crest-derived pharyngeal arch mesenchyme. Dev Biol 255, 230-7.

Jessen WJ, Miller SJ, Jousma E, et al. MEK inhibition exhibits efficacy in human and mouse neurofibromatosis tumors. J Clin Invest 2013:123:340-7.

Jett K, Friedman JM. Clinical and genetic aspects of neurofibromatosis 1. Genetics in medicine: official journal of the American College of Medical Genetics 2010;12:1-11.

Kalinec, G., Nazarali, A. J., Hermouet, S., Xu, N., and Gutkind, J. S. (1992). Mutated alpha subunit of the Gq protein induces malignant transformation in NIH 3T3 cells. Mol Cell Biol 12, 4687-93.

Kirkwood, J.M., L. Bastholt, C. Robert, *et al.* (2012). Phase II, open-label, randomized trial of the MEK1/2 inhibitor selumetinib as monotherapy versus temozolomide in patients with advanced melanoma. *Clin Cancer Res.* 18:555-567.

Kwon CH, Zhao D, Chen J, Alcantara S, Li Y, Burns DK, et al. Pten haploinsufficiency accelerates formation of high-grade astrocytomas. Cancer Res. 2008;68:3286-94.

Lacouture, M.E., M.J. Anadkat, R.J. Bensadoun, *et al.* (2011). Clinical practice guidelines for the prevention and treatment of EGFR inhibitor-associated dermatologic toxicities. *Support Care Cancer.* 19:1079-1095.

Le Gal, F., E. Gordien, D. Affolabi, *et al.* 2005. Quantification of hepatitis delta virus RNA in serum by consensus real-time PCR indicates different patterns of virological response to interferon therapy in chronically infected patients. J Clin Microbiol. 43:2363-2369.

Luke JL, Ott PA, Shapiro GI. (2014) The biology and clinical development of MEK inhibitors for cancer. *Drugs*. 74(18):2111-28.

MEKINIST [Package insert]. (2013). GlaxoSmithKline. May 2013.

Maertens O, Johnson B, Hollstein P, et al. Elucidating distinct roles for NF1 in melanomagenesis. Cancer Discov 2013;3:338-49.

Version Date: August 19, 2020
(2011) Clinical activity of the

Messersmith, W.A., G.S. Falchook, L.A. Fecher, *et al.* (2011). Clinical activity of the oral MEK1/MEK2 inhibitor GSK1120212 in pancreatic and colorectal cancer. *J Clin Oncol.* 29:Abstract 246.

O'hayre, M., Vazquez-Prado, J., Kufareva, I., Stawiski, E. W., Handel, T. M., Seshagiri, S., and Gutkind, J. S. (2013). The emerging mutational landscape of G proteins and G-protein-coupled receptors in cancer. Nat Rev Cancer 13, 412-24.

Onken, M. D., Worley, L. A., Ehlers, J. P., and Harbour, J. W. (2004). Gene expression profiling in uveal melanoma reveals two molecular classes and predicts metastatic death. Cancer research 64, 7205-9.

Onken, M. D., Worley, L. A., Long, M. D., Duan, S., Council, M. L., Bowcock, A. M., and Harbour, J. W. (2008). Oncogenic mutations in GNAQ occur early in uveal melanoma. Invest Ophthalmol Vis Sci 49, 5230-4.

Parsons D, Jones S, Zhang X, Lin J, Leary R, Angenendt P, et al. An integrated genomic analysis of human glioblastoma multiforme. Science. 2008;321:1807-12.

Patil S, Chamberlain RS. Neoplasms associated with germline and somatic NF1 gene mutations. Oncologist 2012;17:101-16.

Reilly KM, Loisel DA, Bronson RT, McLaughlin ME, Jacks T. Nf1;Trp53 mutant mice develop glioblastoma with evidence of strain-specific effects. Nat Genet. 2000;26:109-13.

Robert, C., Dummer, R., Gutzmer, R., Lorigan, P., Kim, K. B., Nyakas, M., Arance, A., Liszkay, G., Schadendorf, D., Cantarini, M., et al. (2013). Selumetinib plus dacarbazine versus placebo plus dacarbazine as first-line treatment for BRAF-mutant metastatic melanoma: a phase 2 double-blind randomised study. Lancet Oncol 14, 733-40.

Robertson KA, Nalepa G, Yang FC, et al. Imatinib mesylate for plexiform neurofibromas in patients with neurofibromatosis type 1: a phase 2 trial. Lancet Oncol 2012;13:1218-24.

Rosenbaum T, Wimmer K. Neurofibromatosis type 1 (NF1) and Associated Tumors. Klinische Padiatrie 2014.

See WL, Tan IL, Mukherjee J, Nicolaides T, Pieper RO. Sensitivity of glioblastomas to clinically available MEK inhibitors is defined by neurofibromin 1 deficiency. Cancer Res. 2012;72:3350-9.

Thomas L, Mautner VF, Cooper DN, Upadhyaya M. Molecular heterogeneity in malignant peripheral nerve sheath tumors associated with neurofibromatosis type 1. Human genomics 2012;6:18.

Tolcher, A.W., J.C. Bendell, A. Patnaik, *et al.* (2011). A phase lb study of the MEK inhibitor GSK1120212 combined with gemcitabine in patients with solid tumors: Interim results. *J Clin Oncol.* 29:Abstract 278.

- U.S. Food and Drug Administration. (2013). FDA approves two drugs, companion diagnostic test for advanced skin cancer [Press release]. Retrieved from <a href="http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm354199.htm">http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm354199.htm</a>.
- U.S. Food and Drug Administration. (2014). FDA approves Mekinist in combination with Tafinlar for advanced melanoma [Press release]. Retrieved from http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm381159.htm.

Van Raamsdonk, C. D., Bezrookove, V., Green, G., Bauer, J., Gaugler, L., O'brien, J. M., Simpson, E. M., Barsh, G. S., and Bastian, B. C. (2009). Frequent somatic mutations of GNAQ in uveal melanoma and blue naevi. Nature 457, 599-602.

Van Raamsdonk, C. D., Griewank, K. G., Crosby, M. B., Garrido, M. C., Vemula, S., Wiesner, T., Obenauf, A. C., Wackernagel, W., Green, G., Bouvier, N., et al. (2010). Mutations in GNA11 in uveal melanoma. N Engl J Med 363, 2191-9.

Weber, J.S., K.T. Flaherty, J.R. Infante, *et al.* (2012). Updated safety and efficacy results from a phase I/II study of the oral BRAF inhibitor dabrafenib (GSK2118436) combined with the oral MEK 1/2 inhibitor trametinib (GSK1120212) in patients with BRAFi-naïve metastatic melanoma. *J Clin Oncol.* 30:Abstract 8510.

Whittaker SR, Theurillat JP, Van Allen E, et al. A genome-scale RNA interference screen implicates NF1 loss in resistance to RAF inhibition. Cancer Discov 2013;3:350-62.

Widemann B, Marcus L, Fisher M, et al. Phase I study of the MEK1/2 inhibitor selumetinib (AZD6244) hydrogen sulfate in children and young adults with neurofibromatosis type 1 (NF1) and inoperable plexiform neurofibromas (PNs). J Clin Oncol 32:5s, 2014 (suppl; abstr 10018).

Wu, X., Li, J., Zhu, M., Fletcher, J. A., and Hodi, F. S. (2012a). Protein kinase C inhibitor AEB071 targets ocular melanoma harboring GNAQ mutations via effects on the PKC/Erk1/2 and PKC/NF-kappaB pathways. Molecular cancer therapeutics 11, 1905-14.

Wu, X., Zhou, J., Rogers, A. M., Janne, P. A., Benedettini, E., Loda, M., and Hodi, F. S. (2012b). c-Met, epidermal growth factor receptor, and insulin-like growth factor-1 receptor are important for growth in uveal melanoma and independently contribute to migration and metastatic potential. Melanoma Res.

Wu, X., Zhu, M., Fletcher, J. A., Giobbie-Hurder, A., and Hodi, F. S. (2012c). The protein kinase C inhibitor enzastaurin exhibits antitumor activity against uveal melanoma. PloS one 7, e29622.

Yamaguchi, T., R. Kakefuda, N. Tajima, *et al.* (2011). Antitumor activities of JTP-74057 (GSK1120212), a novel MEK1/2 inhibitor, on colorectal cancer cell lines in vitro and in vivo. *Int J Oncol.* 39:23-31.

Yan N, Ricca C, Fletcher J, Glover T, Seizinger BR, Manne V. Farnesyltransferase inhibitors block the neurofibromatosis type I (NF1) malignant phenotype. Cancer Res 1995;55:3569-75.

Yang FC, Ingram DA, Chen S, et al. Nf1-dependent tumors require a microenvironment containing Nf1+/-- and c-kit-dependent bone marrow. Cell 2008;135:437-48.

Zhu Y, Ghosh P, Charnay P, Burns DK, Parada LF. Neurofibromas in NF1: Schwann cell origin and role of tumor environment. Science 2002;296:920-2.

Zhu Y, Guignard F, Zhao D, Liu L, Burns D, Mason R, et al. Early inactivation of p53 tumor suppressor gene cooperating with NF1 loss induces malignant astrocytoma. Cancer Cell. 2005;8:119-30.

Zingone, A., N. Korde, J. Chen, *et al.* (2011). Molecular characterization and clinical correlations of MEK1/2 inhibition (AZD6244) in relapse or refractory multiple myeloma: analysis from a phase II study. *Blood (ASH Annual Meeting Abstracts).* 118:Abstract 306.

## Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol S2: Trametinib/GNAQ/GNA11

### Appendix I

Rev. 12/16, 3/17

### **Patient Pill Calendar**

### **Pill Calendar Directions**

- 1. Take your scheduled dose of each tablet at around the same time each day.
- 2. Please bring the empty bottle or any leftover tablets and your pill calendar to your next clinic visit.
- 3. Take trametinib (GSK1120212) once daily by mouth either 1 hour before or 2 hours after a meal.
- 4. If a dose of trametinib is missed, only make up this missed dose if it is still more than 12 hours until the next scheduled dose.
- 5. Trametinib should be stored at 2-8°C (36-46°F). Refrigerate. Do not freeze.
- 6. Trametinib should not be crushed, dissolved, or chewed.
- 7. Do not take an additional dose as a replacement if vomiting were to occur after a dose of trametinib.

### **Patient Pill Calendar**

This is a calendar on which you are to record the time and number of tablets you take each day. You should take your scheduled dose of each tablet. **Note the times and the number of tablets that you take each day.** If you develop any side effects, please record them and anything you would like to tell the doctor in the space provided. Bring any unused tablets and your completed pill calendar to your doctor's visits.

### **Trametinib**

| | | Date | | Time | Number of | Use the space below to make notes about things you |
|---|---|---|---|---|---|---|
| | | | | tablets | tablets | would like to tell the doctor (including unusual |
| DAY | Month | Day | Year | taken | taken | symptoms you experience, other medicine you have taken and anything else you think would be of interest.) |
| 1 | WOITH | Day | Tear | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| 5 | | + | | | | |
| 6 | | | | | | |
| 7 | | | | | | |
| 8 | | | | | | |
| 9 | | | | | | |
| 10 | | | | | | |
| 11 | | | | | | |
| 12 | | | | | | |
| | | - | | | | |
| 13 | | | | | | |
| 14 | | | | | | |
| 15 | | | | | | |
| 16 | | | | | | |
| 17 | | | | | | |
| 18 | | | | | | |
| 19 | | | | | | |
| 20 | | | | | | |
| 21 | | | | | | |
| 22 | | | | | | |
| 23 | | 1 | | | | |
| 24 | | 1 | | | | |
| 25 | | | | | | |
| 26 | | | | | | |
| 27 | | | | | | |
| 28 | | | | | | |

| Patient Signature: | Date: |
|--------------------|-------|

# Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol S2: Trametinib/GNAQ/GNA11

## Appendix II

| Trametinib Ophthalmi | c Exam Form | | | |
|---|---|---|---|---|
| Please use the form on the following page for docum appropriate to the clinical situation. | enting ophthalmic | exam | nination | is as |
| Subject Name: | | | | |
| Note to examiner: Please assess particularly for washing to the second of the second o | <b>nended</b> For patien | ts in v | whom i | |
| OPHTHALMIC EXAMINATION | | | | |
| 1. Date of Examination: | //<br>dd / mmm / yyyy | | | |
| VISUAL ACUITY | | | | |
| Enter corrected visual acuity | OD: | OS: | | |
| TONOMETRY | | | | |
| Enter IOP (mmHg) | OD: | OS | | |
| INDIRECT FUNDOSCOPY | | | | |
| Indirect Exam: Indicate normal or specify abnormalities | OD: | OS: | | |
| CONFRONTATION VISUAL FIELD EXAM OR AUTOR or 30-2 or equivalent if using a non-Humphrey instru | | Y (e.ç | ı., Hum | phrey 24-2 |
| Indicate normal or specify any abnormalities | OD: | OS | OS: | |
| OPTICAL COHERENCE TOMOGRAPHY (strongly re | commended) | | | |
| Indicate normal or specify any abnormalities | OD: | OS | OS: | |
| COLOR FUNDUS PHOTOS (recommended if retinal | abnormalities are r | noted | )* | |
| Indicate normal or specify any abnormalities | OD: | OS: | | |
| FLORESCEIN ANGIOGRAPHY (suggested if retinal a indicated)* | abnormalities are n | oted | and tes | st clinically |
| Indicate normal or specify any abnormalities | OS: | | | |
| Were any of the following noted on ocular history or exa | | Yes | No | |
| History of CSR? | | | | |
| Evidence of new optic disc cupping? | | | | |
| Evidence of new visual field defects? | | | | |
| EXCLUSION CRITERIA | | | | No |
| <ul> <li>History of RVO?</li> <li>If yes, patient is not eligible for the study.</li> </ul> | | | | |

| <br> | · |
|------|---------------------------------------|

| ECOG-ACRIN | EAY131-S2 |
|-----------------------|-------------------------------|
| Cancer Research Group | Version Date: August 19, 2020 |

Printed Name: \_\_\_\_\_ Date: \_\_\_\_

# Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol S2: Trametinib/GNAQ/GNA11

Rev. Add13 Appendix III

### **Actionable Mutations for Sub-Protocol EAY131-S2**

| Gene Name | Variant ID | Variant Type | Level of Evidence<br>Code | Variant<br>Description |
|---|---|---|---|---|
| GNA11 | COSM52969 | SNV | 2 | p.Q209L |
| GNA11 | COSM52970 | SNV | 2 | p.Q209P |
| GNAQ | COSM28757 | SNV | 2 | p.Q209L |
| GNAQ | COSM28758 | SNV | 2 | p.Q209P |
| GNAQ | COSM28760 | SNV | 2 | p.Q209R |
| GNAQ | COSM52975 | SNV | 3 | p.R183Q |

Other novel GNAQ or GNA11 activating mutations not listed in the above table but identified by one of the designated outside laboratories as described in the MATCH Master Protocol will also be considered actionable mutations (aMOIs) at Level of Evidence Code 3. Please refer to Section 1.4.2 of the MATCH Master Protocol for more information.

# Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol S2: Trametinib/GNAQ/GNA11

## **Appendix IV:**

### **Patient Clinical Trial Wallet Card**

